# PHASE 1 STUDY OF THE SAFETY AND IMMUNOGENICITY OF NA-APR-1 (M74)/ALHYDROGEL® CO-ADMINISTERED WITH NA-GST-1/ALHYDROGEL® IN BRAZILIAN ADULTS

**DMID Protocol Number:** 15-0012

**DMID Funding Mechanism:** NIAID Clinical Trial Implementation Cooperative

Agreement (U01)

Pharmaceutical Support Provided by: Not Applicable

Other Identifying Numbers: IND Sponsor Protocol Number SVI-DBL-01

IND Sponsor: Albert B. Sabin Vaccine Institute

**Principal Investigator:** David Diemert, MD FRCP(C)

Co-Principal Investigator: Rodrigo Correa-Oliveira, PhD

**DMID Scientific Lead:** Gregory Dye, MD

**DMID Medical Monitor:** Soju Chang, MD

**DMID Regulatory Affairs Specialist:** Blossom Smith

Version Number: 5

22 July 2015

#### STATEMENT OF COMPLIANCE

The study will be carried out in accordance with Good Clinical Practice (GCP) as required by the following:

- United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46; 21 CFR Part 50, 21 CFR Part 56, and 21 CFR Part 312)
- ICH E6; 62 Federal Register 25691 (1997)
- Brazilian Resolution N
   <sup>o</sup> 466/12 (replacing Resolution N
   <sup>o</sup> 196/96) on Research Involving Human Subjects
- NIH Clinical Terms of Award

All key personnel (all individuals responsible for the design and conduct of this study) have completed Human Subjects Protection Training.

#### **SIGNATURE PAGE**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable US and Brazilian federal regulations and ICH guidelines.

| Site Inve | estigator: | |
|-----------|------------------------------------|-------|
| Signed: | | Date: |
| | Name: David Diemert, MD | |
| | Title: Principal Investigator | |
| Site Inve | estigator: | |
| Signed: | | Date: |
| Signeu. | Name: Rodrigo Correa-Oliveira, PhD | Date. |
| | <u> </u> | |
| | Title: Co-Principal Investigator | |

# **TABLE OF CONTENTS**

| Sta | atemen | t of Comp | liance | ii |
|---|---|---|---|---|
| Sig | nature | Page | | iii |
| Та | ble of C | Contents | | iv |
| Lis | t of Abl | breviation | S | vii |
| Pro | otocol S | Summary . | | ix |
| 1 | Key R | oles | | 1 |
| 2 | Backg | round Info | ormation and Scientific Rationale | 3 |
| | 2.1 | Backgro | und Information | 3 |
| | | 2.1.1 | Hookworm Infection and Justification for Vaccine Development | 3 |
| | | 2.1.2 | Study Site | 4 |
| | | 2.1.3 | Prior Clinical Experience with Hookworm Vaccines | 5 |
| | | 2.1.4 | The Na-GST-1/Alhydrogel® Hookworm Vaccine | 7 |
| | | 2.1.5 | Immunogenicity Studies with Na-GST-1 | |
| | | 2.1.6 | Clinical Experience with Na-GST-1/Alhydrogel® Hookworm Vaccine | 11 |
| | | 2.1.7 | The Na-APR-1 (M74)/Alhydrogel® Hookworm Vaccine | |
| | | 2.1.8 | Studies of Human Immune Responses to Na-APR-1 in Endemic Areas. | 13 |
| | | 2.1.9 | Clinical Experience with the Na-APR-1 (M74)/Alhydrogel® Hookworm | |
| | | | Vaccine | 13 |
| | | 2.1.10 | Clinical Experience with Aluminum-Based Adjuvants | 14 |
| | | 2.1.11 | Clinical Experience with GLA-AF | 14 |
| | 2.2 | Rational | e | 15 |
| | | 2.2.1 | Rationale for the Study | 15 |
| | | 2.2.2 | Rationale for Doses and Dose Schedule to be Studied | 15 |
| | | 2.2.3 | Clinical Development Plan for the Human Hookworm Vaccine | 16 |
| | 2.3 | Potentia | I Risks and Benefits | 17 |
| | | 2.3.1 | Potential Risks | 17 |
| | | 2.3.2 | Procedures Taken to Minimize Risks | 18 |
| | | 2.3.3 | Known Potential Benefits | 18 |
| 3 | Objec | tives | | 20 |
| | 3.1 | Study O | bjectives | 20 |
| | 3.2 | Study O | utcome Measures | 21 |
| | | 3.2.1 | Primary Outcome Measure | 21 |
| | | 3.2.2 | Secondary Outcome Measures | 21 |
| | | 3.2.3 | Tertiary Outcome Measures | 21 |
| | | 3.2.4 | Exploratory Outcome Measures | 22 |
| 4 | Study | Design | | 23 |
| | 4.1 | Substud | ies (if applicable) | 25 |
| 5 | Study | Enrollmei | nt and Withdrawal | 26 |
| | 5.1 | Subject | Inclusion Criteria | 26 |
| | 5.2 | Subject | Exclusion Criteria | 26 |

| | 5.3 | Treatme | ent Assignment Procedures | 28 |
|---|---|---|---|---|
| | | 5.3.1 | Randomization Procedures | |
| | | 5.3.2 | Masking Procedures | 28 |
| | | 5.3.3 | Reasons for Withdrawal and Discontinuation of Vaccinations | 29 |
| | | 5.3.4 | Handling of Withdrawals | |
| | | 5.3.5 | Termination of Study | |
| 6 | Study | Intervent | ionS/Investigational ProductS | |
| | 6.1 | | roduct Description | |
| | | 6.1.1 | Acquisition | 32 |
| | | 6.1.2 | Formulation, Packaging, and Labeling | 32 |
| | | 6.1.3 | | |
| | 6.2 | Dosage | , Preparation and Administration of Study Intervention/Investigational | |
| | | _ | ct | 33 |
| | 6.3 | | ation of Study Intervention/Investigational Product for a Participant | |
| | 6.4 | | tability Procedures for the Study Intervention/Investigational Product(s) | |
| | 6.5 | | ment of Subject Compliance with Study Intervention/Investigational | |
| | | | ct | 34 |
| | 6.6 | | nitant Medications/Treatments | |
| 7 | Study | Schedule | 9 | 36 |
| | 7.1 | | ng | |
| | 7.2 | | ent/Baseline | |
| | 7.3 | Follow-u | qı. | 37 |
| | 7.4 | | udy Visit | |
| | 7.5 | Early Te | ermination Visit | 40 |
| | 7.6 | Unsche | duled Visit | 40 |
| 8 | Study | Procedui | es/Evaluations | 42 |
| | 8.1 | Clinical | Evaluations | 42 |
| | 8.2 | Laborat | ory Evaluations | 42 |
| | | 8.2.1 | Clinical Laboratory Evaluations | 42 |
| | | 8.2.2 | Special Assays or Procedures | 43 |
| | | 8.2.3 | Specimen Preparation, Handling, and Shipping | 45 |
| 9 | Asses | sment of | Safety | 46 |
| | 9.1 | Specific | ation of Safety Parameters | 46 |
| | 9.2 | Method | s and Timing for Assessing, Recording, and Analyzing Safety Parameter | s46 |
| | | 9.2.1 | Adverse Events | 46 |
| | | 9.2.2 | Reactogenicity | 47 |
| | | 9.2.3 | Serious Adverse Events | 51 |
| | | 9.2.4 | Procedures to be Followed in the Event of Abnormal Laboratory Test | |
| | | | Values or Abnormal Clinical Findings | 51 |
| | 9.3 | Reportir | ng Procedures | 51 |
| | | 9.3.1 | Serious Adverse Events | 51 |
| | | 9.3.2 | Regulatory Reporting for Studies Conducted Under DMID-Sponsored | |
| | | | IND | 50 |

| | | 9.3.3 | Regulatory Reporting for Studies Not Conducted Under | |
|---|---|---|---|---|
| | | | DMID-Sponsored IND | 52 |
| | | 9.3.4 | Adverse Events of Special Interest (AESI) | 52 |
| | | 9.3.5 | Medically-Attended Adverse Events (MAAEs) | 53 |
| | | 9.3.6 | Reporting of Pregnancy | 53 |
| | 9.4 | Type ar | nd Duration of Follow-up of Subjects after Adverse Events | 53 |
| | 9.5 | Halting | Rules | 54 |
| | 9.6 | Safety ( | Oversight | 55 |
| | | 9.6.1 | Independent Safety Monitor (ISM) | 55 |
| | | 9.6.2 | Safety Monitoring Committee (SMC) | 55 |
| 10 | Clinic | cal Monite | oring | |
| | 10.1 | Site M | onitoring Plan | 56 |
| 11 | Statis | stical Cor | nsiderations | 57 |
| | 11.1 | Study | Hypotheses | 57 |
| | 11.2 | Sampl | e Size Considerations | 57 |
| | 11.3 | Planne | ed Interim Analyses | 58 |
| | | 11.3.1 | Safety Review | 58 |
| | | 11.3.2 | 2 Immunogenicity Review | 59 |
| | 11.4 | Final A | Analysis Plan | 59 |
| 12 | Sour | ce Docur | nents and Access to Source Data/Documents | 66 |
| 13 | Qual | ity Contro | ol and Quality Assurance | 67 |
| 14 | Ethic | s/Protect | ion of Human Subjects | 68 |
| | 14.1 | Ethica | l Standard | 68 |
| | 14.2 | Institut | tional Review Boards | 68 |
| | 14.3 | Inform | ed Consent Process | 68 |
| | | 14.3.1 | Informed Consent/Assent Process (in Case of a Minor) | 69 |
| | 14.4 | | sion of Women, Minorities, and Children (Special Populations) | |
| | 14.5 | Subjec | ct Confidentiality | 70 |
| | 14.6 | Study | Discontinuation | 70 |
| | 14.7 | Future | Use of Stored Specimens | 70 |
| 15 | Data | | g and Record Keeping | |
| | 15.1 | | Management Responsibilities | |
| | 15.2 | | Capture Methods | |
| | 15.3 | | of Data | |
| | 15.4 | | g/Reports | |
| | 15.5 | _ | Records Retention | |
| | 15.6 | • | ol Deviations | |
| 16 | Publi | cation Po | olicy | 73 |
| 17 | | | erences | |
| Sun | pleme | nts/Appe | endices | 78 |
| - | • | | fulle of Events | 70 |

#### LIST OF ABBREVIATIONS

AE Adverse Event

AESI Adverse Event of Special Interest

APR-1 Aspartic Protease-1
CBC Complete Blood Count

CPqRR Centro de Pesquisas René Rachou cGMP Current Good Manufacturing Practices

CIOMS Council for International Organizations of Medical Sciences

CRF Case Report Form

DMID Division of Microbiology and Infectious Diseases, NIAID, NIH

ELISA Enzyme linked immunosorbent assay

FDA Food and Drug Administration
FIOCRUZ Foundation Oswaldo Cruz
FWA Federalwide Assurance
GCP Good Clinical Practice

GLA-AF Gluco-Pyranosylphospho-Lipid A Aqueous Formulation

GMP Good Manufacturing Practice
GST-1 Glutathione S-Transferase
HBsAg Hepatitis B surface antigen

HBV Hepatitis B virus

hCG Human choriogonadotropin

HCV Hepatitis C virus

HHVI Human Hookworm Vaccine Initiative HIV Human Immunodeficiency Virus

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonisation IEC Independent or Institutional Ethics Committee

IM Intramuscular

IND Investigational New Drug Application

IPInvestigational ProductIRBInstitutional Review BoardISMIndependent Safety MonitorMAAEMedically-Attended Adverse Event

MedDRA Medical Dictionary for Regulatory Activities

MBC Memory B Cell

MOP Manual of Procedures

N Number (typically refers to subjects)

Na Necator americanus

NIAID National Institute of Allergy and Infectious Diseases, NIH, DHHS

NIH National Institutes of Health

PBMC Peripheral Blood Mononuclear Cell

PI Principal Investigator
QA Quality Assurance
QC Quality Control

SAE Serious Adverse Event

SMC Safety Monitoring Committee SOP Standard Operating Procedure

SVI Sabin Vaccine Institute (Albert B Sabin Vaccine Institute; Sabin)

US United States WBC White Blood Cell

WHO World Health Organization

#### PROTOCOL SUMMARY

Title: Phase 1 Study of the Safety and Immunogenicity of Na-APR-1

(M74)/Alhydrogel<sup>®</sup> Co-administered with Na-GST-1/Alhydrogel<sup>®</sup>

in Brazilian Adults

Phase: 1

**Population:** Healthy male and non-pregnant female volunteers aged 18-45

years, inclusive.

Number of Sites: 1 (Americaninhas Vaccine Center, Minas Gerais, Brazil)

Study Duration: 19 months

Subject Participation

**Duration:** 

13 months

Description of Interventions:

- a) The *Na*-APR-1 (M74) candidate vaccine contains recombinant *Na*-APR-1 (M74) adsorbed onto aluminum hydroxide gel (Alhydrogel<sup>®</sup>) and suspended in a solution containing 10mM imidazole, 150mM sodium chloride and 0.3% Empigen BB, with pH 7.4 ± 0.1. The final concentrations of *Na*-APR-1 (M74) and Alhydrogel<sup>®</sup> in the drug product are 0.1mg/ml and 0.8mg/ml respectively. Doses of 10, 30 and 100 μg *Na*-APR-1 (M74) will be delivered IM to the deltoid by injecting different volumes of the 0.1mg/ml preparation.
- b) The **Na-GST-1** candidate vaccine contains the recombinant Na-GST-1 adsorbed onto Alhydrogel<sup>®</sup> and suspended in a solution containing 10mM imidazole and 10% glucose. The final concentrations of Na-GST-1 and Alhydrogel<sup>®</sup> in the drug product are 0.1mg/ml and 0.8mg/ml respectively. Only one dose of Na-GST-1 will be tested (100μg), at a volume of 1.0ml delivered IM to the deltoid.
- c) Gluco-Pyranosylphospho-Lipid A Aqueous Formulation (GLA-AF) is a Toll-like Receptor-4 agonist. Point-of-injection formulations with this immunostimulant will be prepared immediately prior to vaccination by adding an appropriate volume of GLA-AF to Na-APR-1 (M74) and withdrawing an appropriate volume to administer the desired amount of Na-APR-1 (M74) plus 5µg GLA-AF.
- d) To maintain the study blind by ensuring that all subjects receive two injections at each vaccination point, sterile

normal **saline** (0.9%) for injection will be co-administered to

those subjects randomized to receive *Na*-APR-1 (M74) *without* co-administration of *Na*-GST-1.

#### **Objectives:**

#### **Primary:**

#### Safety

 To evaluate the safety and reactogenicity of three different dose concentrations of Na-APR-1 (M74) adjuvanted with Alhydrogel® or Alhydrogel® plus GLA-AF and administered either with or without Na-GST-1, in healthy Brazilian adults.

#### Secondary:

#### <u>Immunogenicity</u>

 To assess the impact of co-administering Na-APR-1 (M74) and Na-GST-1 on antibody production by measuring the antibody levels to each antigen on study Day 126.

#### **Tertiary:**

#### <u>Immunogenicity</u>

- 1. To assess the impact of co-administration of *Na*-GST-1 on the duration of the antibody responses to *Na*-APR-1 (M74), and vice versa.
- 2. To assess the impact of co-administration of *Na*-GST-1 on the distribution of IgG subclass responses to *Na*-APR-1 (M74) and vice versa.
- 3. To assess the impact of co-administration of *Na*-GST-1 and *Na*-APR-1 (M74) on the functional capacity of vaccine-induced antibodies to neutralize the *in vitro* activity of the native enzymes (*Na*-GST-1 and wild type *Na*-APR-1).
- 4. To assess the impact of co-administration of *Na*-GST-1 and *Na*-APR-1 (M74) on the affinity of the antibody interactions with both recombinant antigens.
- 5. To assess the impact of co-administration of *Na*-GST-1 and *Na*-APR-1 (M74) on the production of memory B cells specific for each antigen.

# Description of Study Design:

Double blind, randomized, controlled, dose-escalation Phase 1 clinical trial in hookworm exposed adults living in the area of Americaninhas, Minas Gerais, Brazil. Subjects will receive three

doses of the assigned vaccine delivered intramuscularly on approximately Days 0, 56, and 112.

Safety will be measured from the time of each study vaccination (Day 0) through 14 days after each study vaccination by the occurrence of solicited injection site and systemic reactogenicity events.

Unsolicited non-serious adverse events (AEs) will be collected from the time of the first study vaccination through approximately 1 month after each study vaccination. New-onset chronic medical conditions and Serious Adverse Events (SAEs) will be collected from the time of the first study vaccination through approximately 9 months after the third study vaccination (final visit). Clinical laboratory evaluations for safety will be performed on venous blood collected approximately 14 days after each vaccination.

Immunogenicity testing will include IgG antibody responses to each vaccine antigen, by an indirect enzyme-linked immunosorbent assay (ELISA) and also by ImmunoCAP, on serum obtained prior to each study vaccination and at time points after each vaccination (see Appendix A); antibody affinity by Surface Plasmon Resonance; functional activity of vaccine-induced antibodies via *in vitro* enzyme neutralization assays; and, antigen-specific memory B cell responses.

Recruitment and enrollment into the study will occur on an ongoing basis, with each group being recruited and vaccinated in sequence.

60 subjects will be enrolled into 6 groups of 10:

The first 20 subjects will be entered into Groups 1 and 2 through open sequential enrollment.

- Group 1 double-blind IP allocation (n=10):
  - 5 subjects will receive 10µg Na-APR-1 (M74) delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 10μg Na-APR-1 (M74)
     delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.
- Group 2 double-blind IP allocation (n=10):
  - 5 subjects will receive 10µg Na-APR-1 (M74) plus 5µg GLA-AF delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 10μg Na-APR-1 (M74) plus
     5μg GLA-AF delivered by IM injection in the deltoid

muscle, with 100µg Na-GST-1 administered to the alternate arm.

The next 20 subjects will be entered into Groups 3 and 4 through open sequential enrollment.

- Group 3 double-blind IP allocation (n=10):
  - 5 subjects will receive 30µg Na-APR-1 (M74) delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 30μg Na-APR-1 (M74)
     delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.
- Group 4 double-blind IP allocation (n=10):
  - 5 subjects will receive 30μg Na-APR-1 (M74) plus 5μg GLA-AF delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 30μg Na-APR-1 (M74) plus 5μg GLA-AF delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.

The final 20 subjects will be entered into Groups 5 and 6 through open sequential enrollment.

- Group 5 double-blind IP allocation (n=10):
  - 5 subjects will receive 100μg Na-APR-1 (M74) delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 100μg Na-APR-1 (M74)
     delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.
- Group 6 double-blind IP allocation (n=10):
  - 5 subjects will receive 100µg Na-APR-1 (M74) plus 5µg GLA-AF delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 100μg Na-APR-1 (M74) plus 5μg GLA-AF delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.

Estimated Time to Complete Enrollment:

3 months

22 SWI

#### Schematic of Study Design:

Group Allocation: Open sequential enrollment

Within Group IP Allocation: Double-blind randomized assignment -----



#### **KEY ROLES** 1

#### Individuals:

#### **Principal Investigator:**

David Diemert, MD FRCP(C), Associate Professor George Washington University Department of Microbiology, Immunology, and Tropical Medicine (GW MITM) Washington, DC, USA Tel: 202-994-2909

Fax: 202-994-2913

Email: ddiemert@gwu.edu

#### **Co-Principal Investigator:**

Rodrgio Correa-Oliveira, PhD Centro de Pesquisas René Rachou (CPqRR) - FIOCRUZ Av. Augusto de Lima 1715, Belo Horizonte, Minas Gerais, Brazil

DMID Medical Monitor: Soju Chang, MD

#### **Local Independent Safety Monitor:**

Christiane Cimini, MD

Téofilo Otoni, Minas Gerais, Brazil E-mail: christiane.cimini@ufvjm.edu.br

#### Institutions:

#### Study Site:

Americaninhas Vaccine Center Americaninhas, Municipality of Novo Oriente Minas Gerais. Brazil

Contact Person: Renata Diniz Phone Number: +55 (33) 3532-7015 E-mail: diniz@cpqrr.fiocruz.br

#### **Clinical Laboratory:**

Laboratório Carlos Chagas Rua Sete de Setembro, 2000 - Centro CEP 35010 - 172

Governador Valadares, Minas Gerais, Brazil

Contact Person: Thiago Mourão

Tel: +55 (33) 3271-2525

Fax Number: 55 (33) 3212-5555

E-mail: thiagomourao@chagasgv.com.br

#### **Immunology Laboratories:**

Laboratório de Imunologia Celular e Molecular Centro de Pesquisas René Rachou (CPqRR) - FIOCRUZ Av. Augusto de Lima 1715, Belo Horizonte, Minas Gerais, Brazil

Contact Person: Fernanda Gambogi

Tel: +55 (31) 3349-7715 Fax: +55 (31) 3295-3115

E-mail: gambogi@cpqrr.fiocruz.br

#### Clinical Immunology Laboratory

Dept. of Microbiology, Immunology and Tropical Medicine School of Medicine and Health Sciences The George Washington University 2300 Eye Street NW, Ross 512 Washington, DC 20037

Contact Person: Jill Brelsford Tel: (202) 994-1409

Fax: (202) 994-2913 E-mail: jillb85@gwu.edu

# 2 BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE

# 2.1 Background Information

#### 2.1.1 Hookworm Infection and Justification for Vaccine Development

There is an urgent need for new tools to control human hookworm infection and to reduce its burden of disease in developing countries. This is especially important for children and women of reproductive age who represent populations that are highly vulnerable to the effects of hookworm disease. Up to 65,000 deaths annually have been attributed to human hookworm infection (1). However, the mortality figures pale in comparison to global disease burden estimates that suggest that hookworm may account for the loss of up to 22 million Disability Adjusted Life Years annually (2). With the exception of malaria, hookworm is the most important parasitic disease of humans.

Human hookworm infection is a soil-transmitted helminth infection caused by the nematode parasites *Necator americanus* and *Ancylostoma duodenale*. It is one of the most common chronic infections of humans, affecting up to 740 million people in the developing nations of the tropics (2). The largest number of cases occurs in impoverished rural areas of sub-Saharan Africa, Southeast Asia, China, and the tropical regions of the Americas. Approximately 3.2 billion people are at risk for hookworm infection in these areas. *N. americanus* is the most common hookworm worldwide, whereas *A. duodenale* is more geographically restricted (3).

Hookworm transmission occurs when skin comes into contact with infective third-stage larvae (L3) in fecally contaminated soil. The L3 have the ability to penetrate the skin, usually of the hands, feet, arms, buttocks and legs. The L3 invade human tissues and enter the gastrointestinal tract where they molt to the adult stage approximately 5-9 weeks following initial host entry. Adult hookworms are approximately 1 cm long parasites that cause host injury by attaching to the mucosa and submucosa of the small intestine to produce intestinal blood loss. There is a direct relationship between hookworm intensity (as determined by fecal egg counts) and host blood loss; typically the presence of between 40 and 160 adult hookworms in the intestine results in blood loss sufficient to cause anemia and malnutrition. The term "hookworm disease" refers primarily to the iron deficiency anemia and protein losses that occur in moderate and heavy infections (4). When host iron stores become depleted, there is a direct correlation between hookworm intensity and reduced host hemoglobin, serum ferritin, and protoporphyrin. Because of their low iron stores, children and women of reproductive age are the populations considered the most vulnerable to hookworm-associated blood loss (4-11).

In children, chronic hookworm infection and the resultant iron deficiency anemia have been shown to impair physical and intellectual development (3, 12, 13). Preschool children are particularly vulnerable to the effects of hookworm anemia and disease (8). In addition to its health impact on children, hookworm infection also affects adults. Unlike other soil-transmitted helminth infections such as ascariasis and trichuriasis, in which the highest intensity infections

•

occur almost exclusively in school-aged children, it has been shown that high-intensity hookworm infections may also occur in adults (14-16).

The primary approach to hookworm control worldwide has been the frequent and periodic mass administration of benzimidazole anthelminthics to school-aged children living in high-prevalence areas. In 2001, the World Health Assembly adopted Resolution 54.19, which urges member states to provide regular anthelminthic treatment to high-risk groups with the target of regular treatment of at least 75% of all at-risk school-aged children. However, cure rates for a single dose of a benzimidazole are sub-optimal, particularly for mebendazole (17-20). These concerns have prompted interest in developing alternative tools for hookworm control (3, 21, 22). Vaccination to prevent the anemia associated with moderate and heavy intensity hookworm infection would alleviate the public health deficiencies of drug treatment alone.

The feasibility of developing a hookworm vaccine is based on the previous success of using live, irradiated hookworm larvae (L3 stage) as a vaccine for canine hookworm infection. This provided the experimental basis for the commercial development of a canine hookworm vaccine, which was marketed in the United States during the early 1970s. However, it is not realistic to develop a live L3 vaccine for humans due to multiple reasons including high production costs, challenging storage requirements, a short shelf life, and a lack of sterilizing immunity.

Alternatively, the strategy being pursued is to identify key hookworm proteins to which protective immune responses are directed in the animal models for this infection (namely the canine model) and to produce these as recombinant proteins that could then be used as vaccine antigens. This effort focused initially on identifying antigens expressed by the invading larvae (L3). In addition, a separate strategy has been to identify targets of the adult stage of the hookworm lifecycle; since hookworms attach onto the intestinal lumen and ingest host blood, antibodies could also be ingested that if directed against key hookworm proteins, would interfere with their function, ultimately resulting in the death or reduced fecundity of the worm.

#### 2.1.2 Study Site

The trial described in this protocol is being conducted to evaluate the safety and immunogenicity of two adult stage *N. americanus* candidate vaccine antigens, and will be conducted in Americaninhas, a town located in the Municipality of Novo Oriente de Minas, 500 km northwest of Belo Horizonte, the capital of the Brazilian state of Minas Gerais. The Brazilian Fundação National de Saúde (National Health Foundation) estimates that there are approximately 1000 people living in the urban municipal center of Americaninhas, with another 4000 living in the surrounding rural areas. The area is hilly and characterized by a tropical altitude climate, with an average temperature of 24°C, and experiences a long rainy season between November and March; annual rainfall is 1300-2000 mm. The majority of inhabitants are involved in rural subsistence farming, growing mainly coffee, manioc and beans. Cattle ranching is another important source of income. Houses are predominantly made from concrete or from a combination of wood and mud and have either tiles or iron sheets for roofing. Only approximately 50% of these homes have a latrine and people commonly collect their water from local springs. There is only one government-run health clinic in the area staffed by one physician (part-time) and two auxiliary health workers who are paid by the municipality.

•

Americaninhas has been chosen as a site for testing hookworm vaccines based on prevalence surveys conducted over the past several years, and the good working relationship that has been established between the research staff, the local health authorities, and the community. Starting in 2004, epidemiological studies have been conducted by the study team in the town of Americaninhas and surrounding areas in order to identify the populations at greatest risk for heavy hookworm infection and to conduct post-treatment hookworm re-infection studies in order to inform the sample size calculations for Phase 1 and Phase 2 studies in the region. These studies have been challenging due to a number of environmental obstacles including the isolation of the region, the hilly terrain, and the large distances between dwellings. Geographic Information System/Remote Sensing identified high levels of vegetation as a critical feature of the infection sites. Overall, the force of infection in Minas Gerais is high. It was estimated that post-treatment hookworm infection occurs in approximately 300 per 1,000 individuals per year, which represents a level of transmission that is comparable to other areas considered to have intense or high transmission, such as in East Africa. The overall prevalence of *N. americanus* hookworm infection is approximately 68 percent, with approximately one-half of the population also infected with Ascaris lumbricoides and with Schistosoma mansoni (23).

Over the past 8 years, a research team based at the Centro de Pesquisas René Rachou (CPqRR) in Belo Horizonte, Minas Gerais, Brazil, has collaborated with researchers at the George Washington University (GWU) and the Sabin Vaccine Institute to develop a major outpatient clinical trial facility in Americaninhas. CPqRR is a member institution of the Fundação Oswaldo Cruz (FIOCRUZ), which is the principal research organization of the Brazilian federal Ministry of Health. CPqRR, with funding from the Sabin Vaccine Institute and the Brazilian federal Ministry of Health, has invested in dedicated clinical facilities for conducting clinical trials of investigational products in the town of Americaninhas. At the field site in Americaninhas, the CPqRR has built a vaccine-testing center in the town for the conduct of vaccine and other clinical trials. To date, two Phase 1 hookworm vaccine trials have successfully been conducted at this site.

The vaccine-testing center in Americaninhas is equipped with basic medical instrumentation and supplies to stabilize and treat acute medical problems. The clinic has an automatic generator back-up electrical supply, in case of loss of municipal power. This clinic consists of an observation room, a waiting room, three clinical examination rooms, a small clinical pharmacy with temperature-monitored refrigerator, a small laboratory and phlebotomy room, a room for treating acute medical problems such as immediate allergic reactions following vaccination, and a secure document storage room. The facilities in Americaninhas have access to emergency care and accommodations in the event of serious or other adverse events that require such management. Americaninhas is located approximately a one-hour drive from the nearest town with a hospital.

#### 2.1.3 Prior Clinical Experience with Hookworm Vaccines

The first hookworm vaccine to be tested in humans was the *Na*-ASP-2 (Ancylostoma Secreted Protein-2 of *N. americanus*) Hookworm Vaccine, consisting of recombinant *Na*-ASP-2 expressed in *Pichia pastoris* and adsorbed to aluminum hydroxide gel (Alhydrogel<sup>®</sup>). *Na*-ASP-2 is an excretory/secretory product produced by infective *N. americanus* larvae upon penetration of human skin. In animal models, vaccination with this recombinant antigen was shown to result in reduced worm burdens after challenge infection. Accordingly, a Phase 1 clinical trial of

several different dose concentrations of the vaccine was conducted in healthy, hookworm-naïve

several different dose concentrations of the vaccine was conducted in healthy, hookworm-naive adults living in the United States, which showed the formulation to be safe, well tolerated and immunogenic (24).

However, upon testing the vaccine in adults who had previously been infected with hookworm in Americaninhas, several volunteers in the lowest dose cohort to be vaccinated developed generalized urticaria within 2 hours of immunization (25). Due to these immediate-type hypersensitivity reactions, vaccinations in this study were halted. Subsequent investigations revealed that the volunteers who developed urticaria upon their first dose of *Na*-ASP-2 had elevated levels of baseline (i.e., pre-vaccination) IgE to the vaccine antigen. Subsequently, a sero-epidemiological survey was conducted in an endemic region of Brazil; this study revealed that even in young children, a significant proportion of individuals have detectable levels of IgE to this protein, likely due to previous infection with *N. americanus* (**Figure 1**). In addition, similar findings were demonstrated for other larval proteins that were being considered as vaccine candidates.

**Figure 1: Anti-Na-ASP-2 IgE antibody levels in residents of a hookworm-endemic region of northeastern Minas Gerais state, Brazil.** Antibody levels were measured by ELISA; each dot represents an individual. Levels are shown for individuals of various age groups, in addition to the 9 participants of the Phase 1 trial of *Na*-ASP-2 in Brazil and the participants of the first Phase 1 trial of *Na*-ASP-2 that was conducted in hookworm-naïve adults in the United States (25).



Due to these cumulative data, clinical development of the *Na*-ASP-2 and other larval-stage antigens as candidate vaccines was halted. Instead, the current strategy is to develop antigens expressed during the adult stage of the hookworm life cycle that play a role in digesting the host hemoglobin that is used by the worm as an energy source. These antigens do not induce

specific IgE antibodies during natural infection, and hence have a low likelihood for inducing allergic reactions upon vaccination.

# 2.1.4 The Na-GST-1/Alhydrogel® Hookworm Vaccine

The nutritional and metabolic requirements of the adult hookworm living in the human intestine are dependent upon degradation of host hemoglobin that has been ingested by the worm. *N. americanus* hookworms depend on host hemoglobin for survival (26). Following hemolysis, adult hookworms use an ordered cascade of hemoglobinases to cleave hemoglobin into smaller molecules (26-31). Aspartic protease-1 of *N. americanus* (*Na*-APR-1) is responsible for initiating the proteolytic cascade in hookworms, as described below (**Section 2.1.7**). After hemoglobin digestion, the freed heme generates toxic oxygen radicals that can be bound and detoxified by molecules such as glutathione S-transferase-1 (GST-1) (32-34). GST-1 of *N. americanus* (*Na*-GST-1) is a critical enzyme that plays a role in parasite blood feeding; used as a vaccine, we hypothesize that the antigen will induce anti-enzyme neutralizing antibodies that will interfere with parasite blood-feeding and cause parasite death or reduce worm fecundity.

Na-GST-1 is a 24-kDa protein with peroxidase enzymatic activity that catalyzes the conjugation of reduced glutathione to a variety of electrophiles (32-34). This hookworm protein belongs to the Nu class of nematode GSTs, which also includes GSTs from the blood-feeding parasite of ruminants, Haemonchus contortus, and the rodent nematode Heligomosoides polygyrus. This class is characterized by diminished peroxidase activity relative to other classes of GSTs, but elevated binding capacity for heme and related products (32, 34-37). X-ray crystallography of Na-GST-1 demonstrates that the protein can form homodimers in solution, which create atypically large binding cavities accessible to a diversity of ligands, including heme (Figure 2) (34). Na-GST-1 binds heme at high affinity in vitro (32, 37). Because both heme and hematin contain oxidative iron, these molecules are potent generators of toxic reactive oxygen species that could potentially damage parasite macromolecules. In vivo, hookworm GSTs may therefore bind and detoxify the heme and hematin byproducts generated during the blood degradation process.

**Figure 2:** Three-dimensional surface plot of *Na*-GST-1. The path to the binding cavity is indicated by the red arrow (34).



Based on their putative role in hookworm blood feeding, both *Na*-GST-1 and its orthologue from the canine hookworm *Ancylostoma caninum* (*Ac*-GST-1) were tested as experimental vaccines in laboratory animals models of infection. In dogs, vaccination with recombinant *Ac*-GST-1 resulted in high levels of antigen-specific antibody (**Figure 3**); following challenge with *A*.

•

caninum infective larvae, significantly lower host worm burdens and fecal egg counts were observed compared to control animals vaccinated only with adjuvant (32). In hamsters, vaccination with recombinant *Ac*-GST-1 also resulted in substantially lower worm burdens (51-54%) following heterologous challenge with *N. americanus* infective larvae compared to controls, as did vaccination with recombinant *Na*-GST-1 followed by homologous larval challenge (32, 33, 38). Because of these encouraging preclinical results, *Na*-GST-1 was manufactured according to current good manufacturing practices (cGMP) and formulated on Alhydrogel® in preparation for clinical trials.

Figure 3: Geometric mean titers of the IgG1 and IgG2 antibody responses of vaccinated dogs against recombinant *Ac*-GST-1 formulated with GlaxoSmithKline's **AS03 adjuvant.** Vaccination time points (1, 2, 3, and 4) and challenge day (C) are marked with arrows (32).



Most importantly, extensive studies have been conducted to test for sensitization to the Na-GST-1 protein in individuals living in a hookworm endemic area who have been repeatedly exposed and infected with N. americanus. As shown in Figure 4, over 1000 individuals of all ages from a hookworm endemic area of Brazil have been tested for serum IgE antibodies to Na-GST-1 using an indirect ELISA. In addition, a subset of these serum samples stratified by age and infection status (n = 179) underwent confirmatory testing at the Johns Hopkins Dermatology, Allergy and Clinical Immunology Reference Laboratory (Baltimore, Maryland) using a custom ImmunoCAP assay. The ImmunoCAP method is considered the standard for measuring specific IgE to antigens in serum. This confirmatory testing demonstrated that none of the samples had Na-GST-1 IqE values above the clinical cut-off of 0.35 kU<sub>4</sub>/L (Figure 5). Therefore, the likelihood of inducing immediate-type hypersensitivity reactions by vaccinating individuals living in hookworm-endemic areas with Na-GST-1 is low and likely not more than that associated with any new vaccine antigen entering clinical trials. The situation with Na-GST-1 is therefore very different from that of Na-ASP-2 in that repeated infection with hookworm does not induce an IgE response to the antigen, most likely due to the fact that it is a protein found in the digestive tract of adult hookworms and is therefore relatively hidden from the

•

human immune system. This lack of antigen-specific IgE in people living in an area of high transmission has served as a major justification for advancing development of *Na*-GST-1 as a candidate vaccine antigen.

Figure 4: Anti-Na-GST-1 IgE levels in (A) adults and children and (B) young children aged 1-10 years (n=128) living in a hookworm-endemic area of Brazil. IgE levels (optical density at 492 nm) were measured by ELISA.

Α.



B. IgE against GST-1 in pediatric population (n=128), 1-10 years old.



Figure 5: Anti-Na-GST-1 IgE levels in a subset of adults and children (n=179) living in a hookworm-endemic area of Brazil. IgE levels (kU<sub>A</sub>/L) were measured by custom ImmunoCAP.



Na-GST-1 has been successfully manufactured and tested in the laboratory and in animals with both Alhydrogel<sup>®</sup> and Alhydrogel<sup>®</sup> plus GLA-AF. Na-GST-1 has been shown to be pure, potent, and stable in both of these two formulations.

The *Na*-GST-1 vaccine formulation to be tested in this study consists of the 24-kDa recombinant protein *Na*-GST-1, adsorbed to an adjuvant, Alhydrogel<sup>®</sup> (aluminum hydroxide suspension) with or without the addition of Gluco-Pyranosylphospho-Lipid A Aqueous Formulation (GLA-AF). The GLA-AF will be added to the Alhydrogel<sup>®</sup> formulation within 24 hours of immunization. The active ingredient is the recombinant *Na*-GST-1 protein that is derived by fermentation of *Pichia pastoris* yeast cells genetically engineered to express *Na*-GST-1.

### 2.1.5 Immunogenicity Studies with Na-GST-1

Several preclinical animal studies have been conducted in both mice and rats to assess the immunogenicity of *Na*-GST-1 in combination with different adjuvants. First, a study conducted in Sprague-Dawley Rats demonstrated that the addition of an adjuvant to recombinant *Na*-GST-1 was necessary, since administration of the recombinant protein without an adjuvant resulted in minimal specific antibody responses.

A second study was conducted in BALB/c mice to assess the effect of co-administering CPG 10104 with recombinant Na-GST-1/Alhydrogel (Figure 8). In this study, mice were vaccinated with Na-GST-1/Alhydrogel at antigen doses ranging from of 0.01 to 31.25  $\mu$ g Na-GST-1 with or without CPG 10104 (5  $\mu$ g) or CPG 10105 (5  $\mu$ g). CPG 10105 is a CpG oligodeoxynucleotide sequence that is similar to CPG 10104 but that is not being proposed to be tested in the study

•

described in this protocol. Mice were vaccinated twice intramuscularly at a 3-week interval, with blood collected for anti-*Na*-GST-1 IgG ELISA two weeks after the second immunization. This study demonstrated a large, highly significant increase in IgG specific for *Na*-GST-1 in the group administered *Na*-GST-1/Alhydrogel<sup>®</sup>/CPG 10104 compared to that administered only *Na*-GST-1/Alhydrogel<sup>®</sup> as shown in **Figure 8**.

Figure 8: Geometric mean anti-*Na*-GST-1 IgG antibody units 2 weeks after the 2<sup>nd</sup> Immunization of BALB/c mice with *Na*-GST-1/Alhydrogel<sup>®</sup> with or without coadministration of CPG 10104 or CPG 10105.



# 2.1.6 Clinical Experience with *Na*-GST-1/Alhydrogel<sup>®</sup> Hookworm Vaccine

The Na-GST-1/Alhydrogel® hookworm vaccine has been tested in two Phase 1 clinical trials in humans in both the United States (n=40) and Brazil (n=102). So far, no significant reactogenicity or safety issues have been observed in these two studies. In study SVI-11-01 in healthy, hookworm-naïve American adults conducted in Washington, DC, 40 volunteers received three vaccinations with up to 100 μg Na-GST-1/Alhydrogel® administered with or without up to 5 μg GLA-AF (NCT01385189). Mild to moderate injection site pain and tenderness were observed in a minority of study subjects; other common adverse events have included mild to moderate headache and nausea. Vaccinations were completed in this study in early January 2014; interim immunogenicity results are currently pending.

The trial in Brazil (SVI-10-01) has tested *Na*-GST-1/Alhydrogel<sup>®</sup> in both hookworm-unexposed (n=36) and hookworm-exposed (n=66) healthy adults (NCT01261130). This study was initiated

•

in Belo Horizonte, a large urban area in the Brazilian state of Minas Gerais, in healthy, hookworm-unexposed adults (n=36) who received up to 100 µg Na-GST-1/Alhydrogel® with or without 2.5 µg GLA-AF. After no significant adverse events were observed in these volunteers, vaccinations were begun at the hookworm-endemic region of Americaninhas in Minas Gerais; this second part of the trial was a randomized, controlled, double-blind study in which subjects received up to 100 µg Na-GST-1/Alhydrogel<sup>®</sup> with or without 2.5 µg GLA-AF (n=60), or the recombinant hepatitis B vaccine (n=6). All volunteers in this study received three intramuscular injections at 0, 2, and 4 months and are being followed for 12 months after the final vaccination. Vaccinations were completed in August 2013 and preliminary immunogenicity results will be available mid 2014. In this study, the Na-GST-1/Alhydrogel® (with or without GLA-AF) appears to be safe and well tolerated in both hookworm-unexposed and hookworm-exposed adults. No vaccine-related SAEs have occurred and the vaccine appears to be well tolerated, with mild-tomoderate injection site pain and tenderness being the most common vaccine-related adverse events. Also, it is important to note that all volunteers who were screened for study SVI-10-01 were tested for IgE antibodies to Na-GST-1: none of these individuals in either Belo Horizonte or Americaninhas had detectable IgE antibodies to the vaccine antigen, as determined by ELISA.

### 2.1.7 The Na-APR-1 (M74)/Alhydrogel® Hookworm Vaccine

As described above, hookworms acquire their nutrition by ingesting blood, lysing the erythrocytes, and digesting the hemoglobin and serum proteins in the gut of the adult worm via a proteolytic cascade (29). Hookworm hemoglobinases have provided efficacy as recombinant subunit vaccines in animal models of hookworm disease, resulting in significant reductions in the intensity of infection and, most importantly, in protection against blood loss (30-32, 37). The Na-GST-1 and Na-APR-1 proteins are both components of the blood-feeding pathway of N. americanus and were selected for clinical development based on their protective efficacy in animal trials. Na-APR-1 is responsible for initiating the proteolytic cascade in N. americanus and catalytically active recombinant APR-1 has been found to confer protection in canine and hamster models of human hookworm disease (29, 31, 37). Vaccinated animals are thought to be protected as a result of induced antibodies that neutralize the catalytic activity of Ac-APR-1 in the gut of the worm (31).

To improve the stability of the recombinant enzyme, two aspartic acid residues were mutated to alanines to make *Na*-APR-1<sub>mut</sub>, which is the same as *Na*-APR-1 (M74), a catalytically inactivated mutant protein. Dogs vaccinated with recombinant *Na*-APR-1<sub>mut</sub> were protected against blood loss and pathology; importantly, animals that were vaccinated with *Na*-APR-1<sub>mut</sub> generated antibodies that neutralized the catalytic activity of wild type *Na*-APR-1 (30). Despite successfully producing large quantities of refolded *Na*-APR-1 and *Na*-APR-1<sub>mut</sub> in *Escherichia coli*, the scalability of protein expression was hampered by issues of yield and aggregation (30). Therefore, as an alternative strategy, recombinant *Na*-APR-1 (M74) is derived by infiltration of *Agrobacterium tumefaciens* strain GV3101, genetically engineered to express *Na*-APR-1 (M74) in *Nicotiana benthamiana* tobacco plants.

The Na-APR-1 (M74)/Alhydrogel<sup>®</sup> vaccine is composed of the 42.18-kDa Na-APR-1 (M74) recombinant protein (0.1 mg/ml of the recombinant protein in 10 mM imidazole, 150 mM sodium chloride and 0.3% Empigen BB, with pH 7.4 ± 0.1), together with 0.8 mg/ml Alhydrogel<sup>®</sup>.

# 2.1.8 Studies of Human Immune Responses to *Na*-APR-1 in Endemic Areas

To assess serologic recognition of *Na*-APR-1<sub>mut</sub> by humans resident in areas of high transmission for *N. americanus*, sera from 648 hookworm-infected individuals from Minas Gerais state, Brazil, were screened for anti-APR-1<sub>mut</sub> antibody responses. Sixty-two percent showed detectable IgG responses (42% had IgG1, 0.6% IgG2, 15% IgG3, 53% IgG4) and only 0.6% had IgE antibodies to *Na*-APR-1<sub>mut</sub> (Table 1). There was no association between the presence of antibody and current infection status (positive or negative), intensity of infection (EPG), or age.

Table 1: Anti-*Na*-APR-1<sub>mut</sub> IgG, IgG subclasses (IgG1-4), IgE, and IgA Antibodies in Brazilian Individuals Living in a Hookworm-Endemic Area.

| ELISA method | lgG1 | lgG2 | IgG3 | IgG4 | Total<br>IgG | IgE | IgA |
|---|---|---|---|---|---|---|---|
| Dichotomous, positive [% (n)] <sup>a</sup> | 42 (270) | 0.6 (4) | 15 (97) | 53 (343) | 62 (401) | 0.6 (4) | 3 (22) |
| Quantitative (µg/ml) <sup>b</sup> | 0.195 ±<br>0.104 | -с | 0.123 ±<br>0.066 | 0.203 ±<br>0.136 | 0.592 ±<br>0.518 | - | - |

<sup>&</sup>lt;sup>a</sup> Positivity as indicated by a reactivity threshold, which was determined from a frequency distribution from the upper 95% CI of the frequency distribution from log<sub>10</sub> transformed OD values from a panel of sera from Brazilian volunteers not resident in an *N. americanus* transmission area (*n*=56) and a panel of control sera from U.S. volunteers (24).

The presence of IgG1 to Na-APR-1 in sera from humans resident in hookworm endemic areas resolves one of the most critical obstacles of gut antigens as targets for vaccines against blood-feeding helminths. Many consider antigens in the gut membrane of blood-feeding nematodes as "hidden," i.e., not continuously presented to the immune system (35). The presence of circulating IgG1 in individuals in Necator endemic areas indicates that natural infection induces a host immune response to Na-APR-1 and that further immunization could augment this existing immune response. Importantly, the immune response to Na-APR-1 is neither of the IgG4 or IgE isotype as seen with other helminth antigens. This might be the result of expression of Na-APR-1 in the host gastrointestinal tract, compared to other organs through which hookworms pass, such as the skin or lung, and bias the immune response toward a T-helper type 2 cytokine profile. Based on the above studies, it is unlikely that Na-APR-1 (M74) will elicit an IgG4 or an IgE antibody response upon vaccination of individuals in high transmission areas, making this vaccine a highly viable hookworm vaccine candidate.

# 2.1.9 Clinical Experience with the *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> Hookworm Vaccine

The Na-APR-1 (M74)/Alhydrogel® Hookworm Vaccine is currently being tested in healthy, hookworm-unexposed adults in a Phase 1 clinical trial taking place in Washington, DC. In this study (SVI-12-01), 40 volunteers are being vaccinated with either 30 μg or 100 μg Na-APR-1 (M74)/Alhydrogel® with or without 2.5 or 5 μg GLA-AF (NCT01717950). Three intramuscular

<sup>&</sup>lt;sup>b</sup> Values are means ± SD. Amounts were not calculated for samples in which <25 individuals were positive for the antibody. <sup>c</sup> Heterologous interpolation of antibody levels to *Na*-APR-1<sub>mut</sub> refers to a calibration scheme in which the calibration curve uses reagents that have a different specificity from those used to measure the analyte of interest; in this case, *Na*-APR-1<sub>mut</sub>-specific antibody ELISA was simultaneously performed alongside a total Ig assay, with the mass values calibrating by interpolating the sample values by the standard curve of the total Ig assay.

vaccinations are being given to each volunteer according to a 0, 2, and 4-month schedule. All study vaccinations were completed in June 2014, with preliminary immunogenicity results available mid 2014. Thus far, there have been no vaccine-related SAEs and related AEs have been limited mostly to mild-to-moderate injection site pain and tenderness.

#### 2.1.10 Clinical Experience with Aluminum-Based Adjuvants

Several licensed vaccines contain aluminum-based adjuvants, including the recombinant hepatitis B vaccine, the tetanus toxoid vaccine, and the diphtheria-tetanus toxoids vaccine.(39, 40) For these aluminum hydroxide-adsorbed vaccines, local reactions such as pain, tenderness, and swelling are experienced in between 7.6% and 16.7% of volunteers in studies that included over 1,200 healthy adults. Fever is seen in 3.2% to 9.3%, headache in 4.1%, and other systemic symptoms such as fatigue, malaise, nausea, and diarrhea at lower frequencies. Urticaria has been reported in 0.1% of individuals vaccinated with the hepatitis B vaccine.

#### 2.1.11 Clinical Experience with GLA-AF

Both Na-GST-1/Alhydrogel® and Na-APR-1 (M74)/Alhydrogel® are being tested in combination with the Toll-like Receptor 4 (TLR4) agonist, Gluco-Pyranosylphospho-Lipid A in Aqueous Formulation (GLA-AF, Infectious Diseases Research Institute [IDRI], Seattle, WA). GLA-AF contains a synthetic monophosphoryl lipid A (MPL) molecule that has TLR4 agonist activity. MPL is itself derived from the lipopolysaccharide (LPS) of Salmonella minnesota, a natural TLR4 agonist that is pyrogenic and can induce toxic shock. LPS, and more specifically, its lipid A component, has long been known for its strong adjuvant effects; however, its high toxicity has precluded its use in a vaccine formulation. Ribi et al showed that the monophosphorylated form of lipid A retains its adjuvant function and almost completely loses its endotoxin effects (41).

There have been many clinical trials involving thousands of subjects in which MPL or a derivative have been administered as vaccine adjuvants to adults and children, including vaccines for human papillomavirus, malaria (42-44), leishmaniasis (45), and hepatitis B (46). In general, these trials have demonstrated that administering MPL to humans is safe and well tolerated; when compared to formulations of vaccine that do not contain MPL, those adjuvanted with MPL may result in a minor increase in the incidence and/or severity of local injection site reactions. However, the addition of MPL also often results in a much improved specific antibody response to the vaccine antigen(s).

Of note, MPL is one of the components of the licensed Cervarix<sup>®</sup> vaccine (GlaxoSmithKline, Research Triangle Park, NC) for the prevention of cervical cancer due to human papillomavirus serotypes 16 and 18. The adjuvant for this vaccine consists of MPL adsorbed to aluminum hydroxide salt and is therefore similar to the combination of GLA-AF and Alhydrogel<sup>®</sup> that we propose testing in combination with *Na*-GST-1 and *Na*-APR-1 (M74) in the study described in this protocol. The Cervarix<sup>®</sup> vaccine has been shown to have a very favorable safety profile after having been tested in tens of thousands of healthy individuals (47, 48).

As mentioned previously, up to 5 µg of GLA-AF has been administered to a small number of human volunteers in combination with both *Na*-GST-1/Alhydrogel<sup>®</sup> and *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup>. In addition, an oil-in-water emulsion of GLA (GLA-SE) has been used in combination with the Fluzone<sup>®</sup> trivalent killed influenza vaccine in a Phase 1 trial. In this study,

doses up to 2.5 µg of GLA-SE were safe and well-tolerated and significantly enhanced influenza-specific antibody responses (49).

#### 2.2 Rationale

### 2.2.1 Rationale for the Study

A product that combines Na-GST-1 and Na-APR-1 (M74) shows promise as an effective bivalent hookworm vaccine because vaccination of laboratory animals with recombinant Na-GST-1 or Na-APR-1 results in significant protection from challenge infections (30, 38). Therefore, vaccination of humans with recombinant Na-GST-1 or Na-APR-1 (M74) holds promise for inducing protection against this infection, particularly the moderate and heavy intensity infections that are associated with clinical sequelae such as intestinal blood loss and iron-deficiency anemia. The Sabin Vaccine Institute has sponsored a series of Phase 1 trials of the Na-GST-1 and Na-APR-1 (M74) candidate antigens in healthy adult volunteers from hookworm endemic areas (Brazil) and non-endemic areas (USA). Given the results of preclinical testing in laboratory animals, it is thought that a vaccine based on a single antigen will not be sufficient to provide adequate protection from disease (50). Instead, the goal is to develop a multi-component vaccine containing at least two recombinant proteins targeting different steps in the hookworm digestion of host hemoglobin. As such, a necessary step in clinical development is to test whether combining Na-GST-1 and Na-APR-1 (M74) results in an increased safety risk or reduced immunogenicity to either antigen, compared to when they are administered individually.

Through the study described in this clinical protocol, we will utilize several state-of-the-art antibody-profiling technologies (see **Section 8.2**) to determine the impact of co-administering the *Na*-GST-1 and *Na*-APR-1 (M74) hookworm vaccines on the immune response to each antigen. In particular, we will compare conventional indirect enzyme-linked immunosorbent assay (ELISA) techniques with cutting-edge antibody and memory B cell immune techniques from other disciplines (e.g., allergy, biotherapy, biodefense etc.) that offer a more comprehensive profiling of the humoral immune response when administering vaccine antigens. This will allow assessment of the humoral immune response during co-administration from several unique perspectives, including memory B cell development, antibody affinity, and antibody function during co-administration and compare them to conventional antibody assays (i.e., ELISA). The introduction of these novel assays early in vaccine clinical development will enable **decision-making on optimal vaccine composition** during clinical development, saving time, expense, and the required number of human research subjects.

#### 2.2.2 Rationale for Doses and Dose Schedule to be Studied

*Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> has not yet been administered to individuals living in a hookworm-endemic area, whereas *Na*-GST-1/Alhydrogel<sup>®</sup> (with or without GLA-AF) has been tested at the same field site as that proposed in the study described in this protocol, in healthy hookworm-exposed adults without any observed safety concerns. Therefore, in the study described in this protocol, *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> will be administered in escalating doses, whereas the dose of *Na*-GST-1/Alhydrogel will be the maximum tolerated dose in the previous studies of this vaccine candidate. Doses of 10, 30 and 100μg of *Na*-APR-1 (M74) were selected for evaluation

based on preclinical studies and to maintain an equal fold-increase in the amount of antigen. The 10µg dose was also selected as the lowest dose for clinical trials due to the difficulty in precisely dispensing lower volumes (both vaccine antigens have been formulated at a protein concentration of 100µg/ml). As mentioned above, selection of the 100µg dose of *Na*-GST-1 is base on preliminary safety and immunogenicity date from the ongoing Phase 1 study of 10, 30 and 100µg *Na*-GST-1 with or without 2.5µg GLA-AF administered to 102 healthy Brazilian adults (protocol SVI-10-01), and the ongoing Phase 1 study of 10, 30, and 100µg of *Na*-GST-1 with or without 1µg or 5µg GLA-AF administered to 40 healthy US adults (protocol SVI-11-01). To date, 100 µg *Na*-GST-1/Alhydrogel administered with 5 µg GLA-AF has been very well tolerated, with no observed vaccine-related Serious Adverse Events and only mild to moderate local injection site pain and tenderness being the most commonly reported adverse events. Unfortunately, the addition of GLA-AF (any dose) to *Na*-GST-1/Alhydrogel did not significantly increase IgG levels to the *Na*-GST-1 antigen. Therefore, GLA-AF will not be tested further in combination with *Na*-GST-1/Alhydrogel.

For the study proposed in this clinical protocol, each subject will be vaccinated three times, on Days 0, 56, and 112. On each vaccination day each subject will receive two injections, one injection per arm. This vaccination schedule was selected to coordinate with the Expanded Program on Immunization as the human hookworm vaccine is intended to target children, including infants. Local subcutaneous nodules, believed to be granulomatous reactions to aluminum hydroxide, have been observed with use of aluminum hydroxide-based adjuvants. Thus, most aluminum hydroxide-adsorbed vaccines are injected intramuscularly (IM) rather than subcutaneously, and intramuscular injection in the deltoid muscle will be used for administration of all investigational products in the study.

#### 2.2.3 Clinical Development Plan for the Human Hookworm Vaccine

The target population for the human hookworm vaccine is children less than 10 years of age living in hookworm endemic areas, since this is the age group that is most at risk of disease from this infection. Prior to conducting clinical trials in this age group, however, both *Na*-GST-1 and *Na*-APR-1 (M74) are being tested in healthy adults living in areas of high hookworm prevalence.

The decision to proceed to Phase 1 testing in children will be taken after the investigators, the Safety Monitoring Committee (SMC), and the Sponsor have reviewed an interim report of the study described in this protocol. This interim report will include the safety and immunogenicity data of <u>all</u> subjects following three immunizations. It is anticipated that the interim report will be available for review in early 2016. Assuming that co-administration of the two antigens in adults does not result in significant safety concerns, testing will proceed to a Phase 1 trial in Brazilian children living in a hookworm endemic area. After safety and immunogenicity of the co-administered products is shown in children, testing of a co-formulated product that contains both *Na*-GST-1 and *Na*-APR-1 (M74) will be started, first in adults and then in children. The dose concentrations and components of the co-formulated product will be determined through the cumulative results of the study described in this protocol and the previous Phase 1 trials of these vaccine antigens.

Besides the vaccine co-administration trial described in this protocol, a second Phase 1 trial to assess the safety and immunogenicity of co-administration of Na-APR-1 (M74) and Na-GST-1

in healthy adults in a hookworm-endemic region of Gabon is also being planned, with anticipated initiation in late 2014. A 0, 28 and 180-day (0, 1 and 6 months) vaccine schedule is being evaluated in the Gabon study, as compared to the 0, 56, and 112-day (0, 2 and 4 months) vaccination schedule evaluated in this protocol. Results from the studies in Gabon and Brazil will be compared to evaluate co-administration safety and immune interference in diverse hookworm-exposed populations, and to decide on antigen doses, formulations, and vaccination schedule to be used in future clinical trials.

The series of Phase 1 trials in adults and children described above will culminate in a large Phase 2 trial in which the co-formulated antigens will be administered to children living in endemic areas. The hookworm vaccine will be compared to a licensed comparator vaccine to evaluate the impact of mean fecal egg counts as well as a variety of clinical and parasitological endpoints. Assuming that an impact on infection is shown in the Phase 2 trial, that there are no new safety issues that arise due to co-formulation of the antigens, and that combining them into one product does not adversely affect the immunogenicity of either, this product will be tested in a pivotal multi-center Phase 3 trial in children. The primary endpoint of the Phase 3 trial will be the incidence of moderate and heavy hookworm infection (as determined by fecal egg counts) following administration of an anthelminthic and vaccination.

#### 2.3 Potential Risks and Benefits

#### 2.3.1 Potential Risks

Risks to subjects are those associated with venipuncture, intramuscular injection of the vaccines, possible reactions to the vaccines, and breach of confidentiality. Risks occasionally associated with venipuncture include pain and bruising at the site of venipuncture, lightheadedness, and syncope (rarely). Intramuscular (IM) injection also may cause transient discomfort and fainting.

Possible local vaccine reactions include pain, swelling, erythema, induration, transient limitation of limb movement, lymphadenopathy, or pruritus at the injection site. Local subcutaneous nodules, believed to be granulomatous reactions to aluminum hydroxide, have been observed with use of aluminum hydroxide-based adjuvants, although these have not been observed with either *Na*-APR-1 (M74)/Alhydrogel® or *Na*-GST-1/Alhydrogel® in the currently ongoing trials of these products. Regardless, most aluminum hydroxide-adsorbed vaccines are injected intramuscularly rather than subcutaneously. Systemic reactions such as fever, headache, malaise, myalgia, and joint pain, may also possibly occur. Immediate hypersensitivity reactions including urticaria, anaphylaxis, or other IgE-mediated responses are possible as with any vaccine. As with any investigational vaccine, there is a theoretical possibility of risks about which we have no present knowledge. Subjects will be informed of any such risks should further data become available.

Phase 1 trials of *Na*-GST-1/Alhydrogel<sup>®</sup> plus GLA-AF and *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> plus GLA-AF have demonstrated similar reactogenicity and safety to either antigen administered without GLA-AF. However, in a study of an influenza vaccine administered with GLA-SE (a formulation similar to GLA-AF), the frequency and intensity of local reactions were greater than when the vaccine was administered without GLA-SE (51).

Female subjects will be cautioned of the unknown risk of the Na-GST-1/Alhydrogel® or Na-APR-1 (M74)/Alhydrogel® vaccines to the fetus. Females of childbearing potential, unless surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), at least 2 years postmenopausal, or practicing abstinence, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner) from 30 days prior to first vaccination until at least one month (defined as 30 days) following the last vaccination. Female subjects will be counseled by a study clinician or nurse, or referred to the local health clinic for evaluation and institution of an appropriate contraceptive method.

#### 2.3.2 Precautions Taken to Minimize Risks

In order to minimize the risk to subjects, all subjects will be monitored closely during their participation in this study. The study vaccines and GLA-AF have been produced according to current Good Manufacturing Practices (GMP) and will be administered by experienced investigators with drugs and equipment available for the treatment of anaphylaxis and other potential adverse reactions. All vaccine doses will be given by intramuscular injection to minimize injection site reactions such as pain. Furthermore, to reduce the likelihood of immediate-type allergic reactions to the vaccine formulations, all potential trial subjects will be screened for detectable IgE antibodies to *Na*-GST-1 and *Na*-APR-1 (M74); individuals with *Na*-GST-1 IgE antibodies detectable by the ELISA assay that are confirmed to be >0.35 kU<sub>A</sub>/L by the ImmunoCAP method will be excluded from participation in the study, as will any individuals with *Na*-APR-1 (M74) IgE antibodies above the ELISA reactivity threshold.

#### **Maintenance of Confidentiality**

Participants will be asked to provide personal health information. All attempts will be made to keep this information confidential within the limits of the law. However, there is a chance that unauthorized persons will see the subjects' personal health information. All records will be kept in a locked file cabinet or maintained in a locked room at the study site. Electronic files will be password protected. Only people who are involved in the conduct, oversight, monitoring, or auditing of this study will be allowed access to the personal health information that is collected. Any publications from this study will not use information that will identify subjects by name.

#### 2.3.3 Known Potential Benefits

Subjects may not receive any direct benefit from participation in this study. It is hoped that information gained in this study will contribute to the development of a safe and effective hookworm vaccine. All subjects will undergo a stool examination for ova and parasites at the Day 140 and Day 380 study visits. Subjects found to have a helminth infection at either of these study visits will be offered appropriate treatment at the conclusion of the study, free-of-charge. Free medical treatment will be provided to all vaccinated subjects during the active immunization phase and the follow-up period. If the investigators judge that a subject requires hospitalization, transportation will be arranged and the medical management of the subject will be monitored by a study physician and the local Independent Safety Monitor. Medical care for ailments not related to vaccination will not extend beyond the study period, but will be referred

to the nearest government-run health clinic. Medical care for ailments related to vaccination will extend at least until the condition has resolved or stabilized (if a chronic condition).

#### 3 OBJECTIVES

### 3.1 Study Objectives

#### **Primary:**

#### Safety

1. To evaluate the safety and reactogenicity of three different dose concentrations of *Na*-APR-1 (M74) adjuvanted with Alhydrogel® or Alhydrogel® plus GLA-AF and administered either with or without *Na*-GST-1, in healthy Brazilian adults.

#### Secondary:

#### **Immunogenicity**

1. To assess the impact of co-administering *Na*-APR-1 (M74) and *Na*-GST-1 on antibody production by measuring the antibody levels to each antigen on study Day 126.

#### Tertiary:

#### <u>Immunogenicity</u>

- 1. To assess the impact of co-administration of *Na*-GST-1 on the duration of the antibody responses to *Na*-APR-1 (M74), and vice versa.
- 2. To assess the impact of co-administration of *Na*-GST-1 on the distribution of IgG subclass responses to *Na*-APR-1 (M74) and vice versa.
- 3. To assess the impact of co-administration of *Na*-GST-1 and *Na*-APR-1 (M74) on the functional capacity of vaccine-induced antibodies to neutralize the *in vitro* activity of the native enzymes (*Na*-GST-1 and wild type *Na*-APR-1).
- 4. To assess the impact of co-administration of *Na*-GST-1 and *Na*-APR-1 (M74) on the affinity of the antibody interactions with both recombinant antigens.
- 5. To assess the impact of co-administration of *Na*-GST-1 and *Na*-APR-1 (M74) on the production of memory B cells specific for each antigen.

#### **Exploratory:**

#### Immunogenicity

1. To assess the cellular immune responses to the *Na*-GST-1 and *Na*-APR-1 (M74) antigens following immunization.

## 3.2 Study Outcome Measures

#### 3.2.1 Primary Outcome Measures

#### Safety

The following parameters will be evaluated for each dose and formulation of *Na*-APR-1 (M74) alone or co-administered with *Na*-GST-1:

- 1. Frequency of solicited injection site and systemic reactogenicity, graded by severity, on the day of each study vaccination through 14 days after each study vaccination.
- 2. Frequency of study vaccine-related serious adverse events from the time of the first study vaccination through approximately 9 months after the last study vaccination.
- 3. Frequency of clinical safety laboratory adverse events.
- 4. Frequency of unsolicited adverse events, graded by severity, from the time of each study vaccination through approximately 1 month after each study vaccination.
- 5. Frequency of new-onset chronic medical conditions through approximately 9 months after the third study vaccination.
- 6. Frequency of Adverse Events of Special Interest through approximately 9 months after the third study vaccination.

### 3.2.2 Secondary Outcome Measures

#### **Immunogenicity**

The following parameters will be evaluated for each dose and formulation of *Na*-APR-1 (M74) alone or co-administered with *Na*-GST-1:

- 1. The IgG level by an indirect enzyme-linked immunosorbent assay (ELISA) on approximately Day 126.
- 2. The IgG level by ImmunoCAP on approximately Day 126.

#### 3.2.3 Tertiary Outcome Measures

#### <u>Immunogenicity</u>

The following parameters will be evaluated for each dose and formulation of *Na*-APR-1 (M74) alone or co-administered with *Na*-GST-1:

1. The IgG antibody response, by an indirect enzyme-linked immunosorbent assay (ELISA) at approximately 7, 14, and 28 days after each vaccination, and approximately 3, 6, and 9 months after the third dose.

- 2. The IgG antibody response, by ImmunoCAP at approximately 7, 14, and 28 days after each vaccination, and approximately 3, 6, and 9 months after the third dose.
- 3. The IgG subclass distribution (IgG1, IgG3, and IgG4) by plate based ImmunoCAP on approximately Day 126.
- 4. The IgG subclass distribution by plate based ImmunoCAP each day of vaccination, approximately 28 days later, and approximately 3 and 6 months after the final vaccination.
- 5. The functional capacity of vaccine-induced antibodies to neutralize the *in vitro* activity of the native enzymes.
- 6. The affinity of the antibody interactions with both recombinant antigens at approximately 7, 14, and 28 days after each vaccination, and 3, 6, and 9 months after the third dose.
- 7. The production of memory B cells specific for each antigen on days of vaccination, approximately 28 days following each vaccination, and 6 and 9 months after the third dose.

#### 3.2.4 Exploratory Outcome Measures

The following parameter will be evaluated for each dose and formulation of *Na*-APR-1 (M74) alone or co-administered with *Na*-GST-1:

1. Cellular immune responses following vaccination.

#### 4 STUDY DESIGN

The study will be conducted as a randomized, placebo-controlled, double-blind Phase 1 dose-escalating clinical trial in healthy adult volunteers living in the hookworm-endemic area of Americaninhas, Brazil.

Prior to beginning study-related activities, the consent and cooperation of local municipal government leaders and representative community members will be sought, after which volunteers will be invited to participate in the study. After providing written informed consent and passing the informed consent comprehension questionnaire, volunteers will undergo eligibility screening, including a complete medical history, physical examination, hematology testing, serum glucose testing, liver and renal function testing, HIV antibody testing, Hepatitis B and C serology, and urinalysis; urine pregnancy testing will be performed on all female volunteers. In addition, all volunteers will be tested for serum IgE antibodies to *Na*-APR-1 (M74) and *Na*-GST-1, and a fecal examination will be performed for ova and parasites. All clinically significant abnormalities will be reviewed with volunteers and referral for follow-up care will be provided. After screening, those volunteers determined to be eligible, based on the inclusion and exclusion criteria, will be invited to participate in the study.

Sixty volunteers will be progressively enrolled into 1 of 6 Groups over a projected 3-month enrollment period, with each subject followed for 13 months post-enrollment (to Study Day 380). Group enrollment will be done in an open sequential fashion, whereas within each Group, investigational product (IP) assignment and vaccination will be done in a randomized double-blind fashion.

The first 20 subjects will be entered into Groups 1 and 2

- Group 1 double-blind IP assignment (n=10):
  - 5 subjects will receive 10μg Na-APR-1 (M74) delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 10μg Na-APR-1 (M74) delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.
- Group 2 double-blind IP assignment (n=10):
  - 5 subjects will receive 10μg Na-APR-1 (M74) plus 5μg GLA-AF delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 10μg Na-APR-1 (M74) plus 5μg GLA-AF delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.

The next 20 subjects will be entered into Groups 3 and 4

- Group 3 double-blind IP assignment (n=10):
  - 5 subjects will receive 30µg Na-APR-1 (M74) delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 30μg Na-APR-1 (M74) delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.
## Group 4 double-blind IP allocation (n=10):

- 5 subjects will receive 30μg Na-APR-1 (M74) plus 5μg GLA-AF delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
- 5 subjects will receive 30μg Na-APR-1 (M74) plus 5μg GLA-AF delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.

The final 20 subjects will be entered into Groups 5 and 6

- Group 5 double-blind IP allocation (n=10):
  - 5 subjects will receive 100μg Na-APR-1 (M74) delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 100μg Na-APR-1 (M74) delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.
- Group 6 double-blind IP allocation (n=10):
  - 5 subjects will receive 100μg Na-APR-1 (M74) plus 5μg GLA-AF delivered by IM injection in the deltoid muscle, with sterile saline administered to the alternate arm.
  - 5 subjects will receive 100μg Na-APR-1 (M74) plus 5μg GLA-AF delivered by IM injection in the deltoid muscle, with 100μg Na-GST-1 administered to the alternate arm.

As with other aluminum hydroxide-adsorbed vaccines, hypersensitivity reactions would be expected to occur within the first 24 hours after receipt of either of the two vaccines, and other severe local or systemic reactions within 72 hours of vaccination. Subjects will therefore be observed for immediate reactions following each vaccination for at least 1 hour, and will have a clinical assessment either in their home or at the study clinic on Days 1, 3, 7, and 14 following each vaccination. See **Appendix A** for the schedule of clinical and laboratory evaluations.

In order to review safety data at each dose of *Na*-APR-1 (M74)/Alhydrogel® prior to testing it in combination with the point-of injection addition of GLA-AF, and to review safety data at each dose of *Na*-APR-1 (M74)/Alhydrogel® prior to dose escalation, Groups will be enrolled and vaccinated in a staggered fashion. Conference calls between the investigators and the Safety Monitoring Committee (SMC) will be scheduled within the week prior to beginning vaccinations in Groups 3 and 5. A cumulative safety report will be submitted to the SMC before beginning vaccinations in these Groups that will include safety data from at least the first 14 days after vaccination of all subjects in the preceding Group. Written approval (via fax or email) to proceed to vaccinations of Groups 3 and 5 must be obtained from the SMC.

The SMC and Independent Safety Monitor will have access to the randomization code for the study, as they may wish to review the data in an unblinded fashion should significant safety questions arise prior to the final unblinding. The trial will <u>not</u> proceed to the next dose Group if any of the stopping criteria listed in **Section 9.5** are met or, in the clinical judgment of the SMC, Independent Safety Monitor, and/or DMID Medical Monitor the next higher dose would pose an unacceptable safety risk to the subjects.

## 4.1 Substudies (if applicable)

Not Applicable.

## 5 STUDY ENROLLMENT AND WITHDRAWAL

Only subjects who meet all of the inclusion and none of the exclusion criteria will be eligible for enrollment into this study. No exemptions will be granted.

A total of 60 subjects will be enrolled. The study population will be enrolled from in and around Americaninhas, a town located in the Municipality of Novo Oriente de Minas, 500 km northwest of Belo Horizonte, the capital of the Brazilian state of Minas Gerais.

Volunteers agreeing to participate will first provide written informed consent and take a true/false comprehension questionnaire. The questionnaire will be administered orally in the case of illiterate volunteers, and for both written and oral questionnaires study staff will use incorrect answers to identify aspects of the study that require clarification and focus on those areas of the informed consent form for further review with the volunteer. All questionnaire questions must be answered correctly, and the informed consent form signed, prior to study screening and enrollment. Volunteers unable to read will place an imprint of their finger in the place of a signature; in addition, an independent witness, who is not a member of the study team, will sign the consent form to attest that the informed consent form was read to the volunteer, the volunteer's questions were answered, and the volunteer answered all comprehension questions correctly. The original signed informed consent form for each volunteer will be maintained as part of that volunteer's study records. A copy of the informed consent form will be provided to every volunteer.

Screening can occur up to 90 days prior to enrollment; enrollment/randomization, and administration of first dose of study products will occur on the same day.

## 5.1 Subject Inclusion Criteria

- 1. Males or non-pregnant females between 18 and 45 years, inclusive.
- 2. Good general health as determined by means of the screening procedure.
- 3. Available for the duration of individual subject study participation (13 months).
- 4. Willingness to participate in the study as evidenced by signing the informed consent document.

## 5.2 Subject Exclusion Criteria

- 1. Pregnancy as determined by a positive urine hCG (if female).
- Subject unwilling to use reliable contraception (as described in Section 2.3.1) from 30 days prior to the first immunization and up until one month following the third immunization (if female and not surgically sterile, abstinent or at least 2 years postmenopausal, or determined otherwise by medical evaluation to be sterile).
- 3. Currently lactating and breast-feeding (if female).
- 4. Inability to correctly answer all questions on the informed consent comprehension questionnaire.

- 5. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies (a history of essential hypertension that is well controlled by medication will not be considered exclusionary.)
- 6. Has a diagnosis of schizophrenia, bipolar disease or other major psychiatric condition that would make compliance with study visits/procedures difficult (e.g., subject with psychoses or history of suicide attempt or gesture in the 3 years before study entry, ongoing risk for suicide).
- 7. Known or suspected immunodeficiency.
- 8. Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
- 9. Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than trace protein or blood on urine dipstick testing with the exception of greater than trace blood detected in females during menses).
- 10. Laboratory evidence of hematologic disease (absolute leukocyte count <3200/mm<sup>3</sup>; absolute leukocyte count >10.8 x 10<sup>3</sup>/mm<sup>3</sup>; hemoglobin <11.4 g/dl [females] or <12.1 g/dl [males]; or, platelet count <130,000/mm<sup>3</sup>).
- 11. Serum glucose (random) greater than 1.2-times the upper reference limit.
- 12. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
- 13. Participation in another investigational vaccine or drug trial within 30 days of starting this study.
- 14. Previous receipt of the Na-GST-1/Alhydrogel® hookworm vaccine.
- 15. Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
- 16. History of a severe allergic reaction or anaphylaxis.
- 17. Severe asthma as defined by the need for daily use of inhalers or emergency clinic visit or hospitalization within the last 6 months.
- 18. Positive test for hepatitis B surface antigen (HBsAg).
- 19. Positive confirmatory test for HIV infection.
- 20. Positive confirmatory test for hepatitis C virus (HCV) infection.
- 21. Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of the volunteer's expected first vaccination in this study or planned use up to one month following the last vaccination.
- 22. Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to the volunteer's expected first vaccination in the study.
- 23. History of a surgical splenectomy.
- 24. Receipt of blood products within the past 6 months.
- 25. Anti-Na-GST-1 IgE antibody level above 0.35 kU<sub>A</sub>/L by the ImmunoCAP method.
- 26. Anti-Na-APR-1 IgE antibody level above ELISA reactivity threshold.

5.3 Treatment Assignment Procedures

#### 5.3.1 Randomization Procedures

Eligible volunteers will be asked to come to the clinic on their scheduled day of enrollment into the study (Day 0). If required, transportation to the clinic will be provided free-of-charge. One or 2 additional eligible volunteers above the number to be enrolled into a given Group may be scheduled as Day 0 visit alternates, if possible. After undergoing a clinical interview and physical examination to ensure that they remain eligible for participation in the study, that they have had blood collected for safety clinical laboratory and baseline immunogenicity assessments, and that females have had a urine pregnancy test performed that is documented to be negative, volunteers will be randomized and enrolled in the order that they present for vaccination.

Within each group, randomization will be done through use of a randomization code, furnished to the study vaccine manager by the data management center. Access to the randomization list will be exclusively limited to the study vaccine manager and assistant. Between vaccination days, the randomization list will be stored in a locked cabinet. The study vaccine manager and assistant will be unblinded, but will not be involved in further evaluation of study subjects or assessment of adverse events. Volunteers will not be considered enrolled in the study until they have received their first dose of vaccine. In the event that a volunteer is randomized but not enrolled on the day of first vaccination, they will be replaced with an eligible alternate. Enrolled subjects that leave the study for any reason following first vaccination will not be replaced. Any alternates not vaccinated will be invited to participate as members of the next Group. Any Group 6 alternates not vaccinated, and therefore not enrolled in the study, will be offered vaccination with a non-study, licensed vaccine such as the tetanus toxoid or influenza vaccine.

## 5.3.2 Masking Procedures

Due to the staggered, dose-escalation design of the trial, it will not be possible to blind to *Na*-APR-1 (M74)/Alhydrogel® dose assignment or GLA-AF co-administration assignment. That is, those subjects enrolled into Group 1 will receive either 10µg *Na*-APR-1 (M74)/Alhydrogel® administered to one arm and sterile saline administered to the alternate arm, or 10µg *Na*-APR-1 (M74)/Alhydrogel® in one arm and 100µg *Na*-GST-1/Alhydrogel® administered to the alternate arm. Subjects enrolled into Group 2 will receive either 10µg *Na*-APR-1 (M74) /Alhydrogel® plus 5µg GLA-AF administered to one arm and sterile saline administered to the alternate arm, or 10µg *Na*-APR-1 (M74) /Alhydrogel® plus 5µg GLA-AF in one arm and 100µg *Na*-GST-1/Alhydrogel® administered to the alternate arm, and so on.

Investigators and subjects will be blinded to the within-Group random allocation to receive co-administered sterile saline or *Na*-GST-1/Alhydrogel<sup>®</sup> until all subjects have completed their Day 140 visit, the safety and secondary immunogenicity outcomes (i.e., anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) IgG antibody results by ELISA) have been monitored and entered into the database, and the database has been "soft-locked" for interim analysis. Procedures to maintain blinding include administering two injections to all subjects at each vaccination point. For this, sterile saline will be co-administered to those subjects randomized to receive *Na*-APR-1 (M74) without co-administration of *Na*-GST-1.

The study vaccine manager will also prepare all investigational product doses (vaccine or sterile saline placebo) in a separate room, and will hand filled syringes to the vaccinator(s). Since the 10 and 30µg doses of the *Na*-APR-1 (M74) formulations are of different volumes (0.1 and 0.3ml, respectively for administration without GLA-AF) than that of *Na*-GST-1, the contents of all syringes will be disguised using opaque tape. As a further precaution, the vaccinator(s) will not be involved in assessments of reactogenicity or adverse events.

Investigators will be unblinded after all subjects have had their study Day 140 visit. After this point, the study will be single-blinded (i.e., subjects will remain blinded to what products they received). The principal justification for unblinding the investigators before the final study visit has been completed is that the safety and immunogenicity data acquired during the vaccination phase of the study will be crucial in guiding the human hookworm vaccine clinical development plan, and we feel that to make an informed decision as to whether or not to proceed to pediatric trials, we must first assess the unblinded data in a timely fashion.

#### 5.3.3 Reasons for Withdrawal and Discontinuation of Vaccinations

Subjects are free to withdraw from the study at any time and for any reason. Subjects who have received vaccine, regardless of the number of doses received, or who developed an AE or SAE will be encouraged to remain in the study to be followed for safety purposes.

Subjects may voluntarily withdraw their consent for study participation at any time and for any reason, without penalty.

A subject may withdraw or be withdrawn from the study for any of the following reasons:

- Medical disease or condition, or any new clinical findings for which continued
  participation, in the opinion of the Principal Investigator or appropriate co-investigator,
  would compromise the safety of the subject, or would interfere with the subject's
  successful completion of the study, or would interfere with the evaluation of responses.
- Subject no longer meets eligibility criteria.
- As deemed necessary by the Principal Investigator or appropriate co-investigator for noncompliance or other reasons.
- Subject withdrawal of consent.
- Subject lost to follow-up.
- Termination of the study.
- New information becomes available that makes further participation unsafe.

The second or third study vaccination may <u>not</u> be administered to a subject if any of the following criteria are met:

- Medical condition (including pregnancy) for which continued participation, in the opinion
  of the Principal Investigator or appropriate co-investigator, would pose a risk to the
  subject or would be likely to confound interpretation of the results.
- Presence of signs or symptoms that could confound or confuse assessment of study vaccine reactogenicity. For subjects with injection site or systemic signs or symptoms, or with an acute illness, including an oral temperature greater than 38.0°C, the study vaccination should/may be postponed/deferred until signs, symptoms, or acute illness have resolved and if within the acceptable protocol-specified window for that visit. If outside this window, the Sponsor must first approve the second or third study vaccination and the documentation of approval should be filed in the subject's chart.
- Any unresolved or continuing solicited or unsolicited Grade 3 adverse event. An
  unresolved or continuing Grade 1 or Grade 2 adverse event is permissible unless, in the
  opinion of the Principal Investigator or appropriate co-investigator, it would render study
  vaccination unsafe or interfere with the evaluation of responses.
- Grade 3 clinical safety laboratory value that does not decrease to Grade 2 or less prior
  to the second or third study vaccination. Any clinical safety laboratory parameter may be
  re-evaluated only once at the central (clinical) laboratory prior to the second or third
  study vaccination. If the clinical safety laboratory value decreases to Grade 2 or less, the
  subject may receive the second or third study vaccination. The second or third study
  vaccination should be scheduled to occur within the acceptable protocol-specified
  window for that visit. If outside this window, the Sponsor must first approve the study
  vaccination and the documentation of approval should be filed in the subject's chart.
- Severe or sustained reaction or disability related to the first study vaccination.
- New onset of illness or condition that meets exclusion criteria.
- Subject no longer meets eligibility criteria.
- As deemed necessary by the Principal Investigator or appropriate co-investigator for noncompliance or other reasons.
- Subject refusal of further study vaccination.
- Subject withdrawal of consent.
- Subject lost to follow-up.
- Termination of the study.
- New information becomes available that makes further participation unsafe.

## 5.3.4 Handling of Withdrawals

The primary reason for withdrawal from the study will be recorded on the appropriate data collection form. Subjects will be encouraged to complete the Early Termination Visit. The Early Termination Visit procedures are listed in **Section 7.5**. Although subjects are free to withdraw at any time or may be withdrawn by the Principal Investigator or appropriate co-investigator at any time, subjects who receive at least one dose of study vaccines will be encouraged to remain in the study for follow-up safety assessments and collection of venous blood samples for immunogenicity testing. Every attempt will be made to follow all adverse events, including solicited injection site and systemic reactions, serious adverse events, and new-onset chronic medical conditions ongoing at the time of early withdrawal to resolution.

In the case of subjects who fail to appear for a follow-up safety assessment, extensive effort (i.e., three documented contact attempts via in-person visits to the subject's home, made on separate occasions) will be made to locate or recall them, or at least to determine their health status. These efforts will be documented in the subject's records.

## 5.3.5 Termination of Study

If a dose of vaccine is considered significantly reactogenic (see Section 9.2.2), dose escalation and/or additional vaccinations will be suspended until reviewed by the Independent Safety Monitor, SMC, and study sponsor. Any recommendation of the Independent Safety Monitor, DMID Medical Monitor, and SMC to resume or suspend further injections (either for an individual subject or an entire dose Group) will be communicated in writing to the sponsor and Principal Investigator. All communications from the SMC will subsequently be forwarded by the investigators to the applicable IRBs.

## 6 STUDY INTERVENTIONS/INVESTIGATIONAL PRODUCTS

Investigators will receive the current versions of the Clinical Investigator's Brochures for *Na*-GST-1/Alhydrogel® and *Na*-APR-1 (M74)/Alhydrogel®, which comprehensively describe all available preclinical and human experience with the experimental vaccines. If relevant new information becomes available during the course of the trial, the investigators will receive the revised Investigator's Brochure(s).

## 6.1 Study Product Description

## 6.1.1 Acquisition

Vials of *Na*-GST-1/Alhydrogel<sup>®</sup>, *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup>, GLA-AF, and sterile saline for injection for this study will be supplied to the study site by the Sabin Vaccine Institute. *Na*-GST-1/Alhydrogel<sup>®</sup>, *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup>, GLA-AF, and the sterile saline placebo will be transported to the study site at 0.5°C to 10°C; temperature recording devices will accompany the vaccines at all times during transport to ensure temperature limits have not been violated.

## 6.1.2 Formulation, Packaging, and Labeling

## 6.1.2.1 Na-APR-1 (M74)/Alhydrogel®

*Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> is supplied as a sterile milky-white suspension (when shaken slightly). Each 2.0 ml vial contains a 0.1 mg/ml suspension of *Na*-APR-1 (M74) adsorbed to 0.8 mg/mL of Alhydrogel<sup>®</sup> in a solution containing 10 mM imidazole, 150 mM sodium chloride and 0.3% Empigen BB, with pH 7.4 ± 0.1. The maximum dose that will be administered is 100 μg of *Na*-APR-1 (M74), or 1.0 ml of the final drug product. This volume contains the equivalent of approximately 400 μg aluminum. Lower doses of *Na*-APR-1 (M74) are delivered by injecting smaller volumes of the 0.1 mg/ml suspension: for example, 0.3 ml will be injected to deliver 30 μg *Na*-APR-1 (M74). For all doses, the ratio of *Na*-APR-1 (M74) to Alhydrogel<sup>®</sup> will therefore remain constant: for the 30 and 100 μg doses of *Na*-APR-1 (M74) the respective amounts of Alhydrogel<sup>®</sup> will be 240 and 800 μg (corresponding to approximately 120 and 400 μg aluminum, respectively). *Na*-APR-1 (M74) protein expression was completed at Fraunhofer Center for Molecular Biotechnology (FhCMB/Newark, DE) and purification and vialing at the Walter Reed Army Institute of Research (WRAIR/Silver Spring, MD). The product conforms to established requirements of purity, sterility, safety, and identity.

## 6.1.2.2 Na-GST-1/Alhydrogel®

Na-GST-1/Alhydrogel<sup>®</sup> is supplied as a sterile milky-white suspension (when shaken slightly). Each 2.0 ml vial contains 1.35 ml of a 0.1 mg/ml suspension of Na-GST-1 adsorbed to 0.8 mg/ml of Alhydrogel<sup>®</sup> in a buffer consisting of 10% glucose and 10 mM imidazole, pH 7.4.

Glucose acts as an excipient and imidazole as the buffer based on evidence that these components specifically enhance the stability and solubility of *Na*-GST-1. The dose that will be administered in this study is 100 µg of *Na*-GST-1, or 1.0 ml of the final drug product. This volume contains the equivalent of approximately 400µg aluminum. *Na*-GST-1/Alhydrogel<sup>®</sup> was manufactured, formulated and vialed at Aeras Global Vaccine Foundation (Rockville, Maryland, USA).

## 6.1.2.3 Glucopyranosyl-Lipid A Aqueous Formulation (GLA-AF)

GLA-AF will be supplied to the trial site as a 0.5 mL aqueous solution in multi-dose vials containing 25 µg/mL of GLA without preservative. Appropriate volumes of GLA-AF will be withdrawn from the multi-dose vials using a syringe and added to a vial containing *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup>, or vice versa (described in the Investigator's Brochure). The mixture must be administered not more than 24 hours after mixing the GLA-AF with *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup>.

#### 6.1.2.4 Saline Placebo

Sterile isotonic (0.9%) sodium chloride solution ("normal saline") for injection, U.S. Pharmacopeia (USP), will be procured and shipped to the study site at ambient temperature. Normal saline is a clear liquid. In study subjects randomized to receive *Na*-APR-1 (M74) without co-administered *Na*-GST-1, normal saline will be administered intramuscularly as placebo in an equal volume to the *Na*-APR-1 (M74). It will be administered in the deltoid muscle of the arm opposite to the one in which the *Na*-APR-1 (M74) is delivered so that all study subjects receive two injections on each day of vaccination, thus maintaining the study blind.

#### 6.1.3 Product Storage and Stability

Vaccines, GLA-AF, and placebo will be stored at the site in a refrigerator at 2°C to 8°C until just prior to administration and will <u>not</u> be frozen; refrigerator temperature will be monitored continuously. All vaccine vials will be stored in the upright position.

## 6.2 Dosage, Preparation and Administration of Study Intervention/Investigational Product

Doses of *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> and *Na*-GST-1/Alhydrogel<sup>®</sup> administered without GLA-AF will be prepared by withdrawing appropriate volumes into syringes of appropriate size. The *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> plus GLA-AF formulations will be prepared by adding appropriate volumes of GLA-AF solution to vials of *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup>, or vice versa, within 24 hours of vaccination. Doses of the sterile saline control will be prepared by withdrawing the appropriate volume into syringes of appropriate size.

Vaccine doses will be administered by qualified study personnel (a study nurse or physician) in the deltoid muscle of the appropriate arm after disinfecting the skin with an alcohol swab and allowing it to dry.

# 6.3 Modification of Study Intervention/Investigational Product for a Participant

There will be no dose modifications. If a subject's second and/or third dose of study vaccination is deferred, it should be rescheduled to occur within the acceptable protocol-specified window for that visit. If this period elapses, the site must obtain prior approval from the Sponsor to administer the second and/or third study vaccination and the documentation of approval should be filed in the subject's chart. Subjects who do not receive the second and/or third study vaccination will be asked to return for safety assessments and for scheduled venous blood sample collections for immunogenicity testing and will be followed for the duration of the study.

Unblinding can occur upon request of the Independent Safety Monitor or the SMC at any time during the study.

# 6.4 Accountability Procedures for the Study Intervention/Investigational Product(s)

Study vaccines, GLA-AF, and sterile saline placebo supplies must be received by a designated person at the study site, handled and stored safely and properly, and kept in a secure location to which only the designated individuals have access. Study-site personnel are responsible for maintaining accurate records of the vaccine supplies (i.e., *Na*-GST-1/Alhydrogel<sup>®</sup>, *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup>, the sterile saline placebo, and GLA-AF) received, the quantities administered to study subjects, and the amounts remaining at the conclusion of the study.

After administration of vaccine or GLA-AF doses, the empty or wasted vials will be accounted for and stored at the study site until monitoring by the study Sponsor or their designee. At the conclusion of the study, all used and unused *Na*-GST-1/Alhydrogel<sup>®</sup>, *Na*-APR-1 (M74) /Alhydrogel<sup>®</sup>, and GLA-AF vials will be returned to the Sponsor or destroyed on site upon direction from the Sponsor, or maintained at 2 to 8°C until further notice from the Sponsor regarding their disposition.

# 6.5 Assessment of Subject Compliance with Study Intervention/Investigational Product

Not Applicable.

## 6.6 Concomitant Medications/Treatments

Administration of any medications, therapies, or vaccines will be recorded on the appropriate data collection form. Concomitant medications will include all medications taken within the 30 days prior to enrollment, 28 days after each dose of study product, and for new-onset chronic medical conditions through the end of participation in the study for each subject. Prescription and over-the-counter drugs will be included as well as vitamins and supplements.

Use of new medication will prompt an evaluation for the presence of a new diagnosis of chronic medical disease or chronic medical condition.

Medications that might interfere with the evaluation of the investigational product should not be used unless absolutely necessary. Medications in this category include, but are not limited to, glucocorticoids, i.e., high dose oral, parenteral and daily inhaled steroids, and immunosuppressive or cytotoxic drugs. Other than from participation in this study, subjects should not receive experimental agents, including vaccines, for the duration of the study.

The administration of licensed vaccines, should be delayed until 28 days after the last administration of the investigational vaccine.

\_\_\_\_\_

## 7 STUDY SCHEDULE

The following sections provide a detailed listing of the procedures and tests to be performed in this study at designated time points. The total volume of blood (approximately 669 mL) to be collected from each volunteer over their 13-month participation in the trial is approximately the volume collected when donating one unit of blood and should not compromise the health of trial subjects. See **Appendix A** for the schedule of study procedures.

## 7.1 Screening

The following procedures will be performed upon initial screening (note that all procedures might not be performed on the same day):

- 1. Explain the study and Informed Consent to the volunteer.
- 2. Ensure the subject has passed the informed consent comprehension questionnaire, has signed the Informed Consent and receives a signed copy of the Informed Consent.
- 3. Elicit a complete medical history, including medication history, and for female subjects, a menstrual and contraceptive history and/or history of surgical sterility.
- 4. Administer a physical examination, including vital signs (heart rate, respiratory rate, arterial blood pressure, and oral temperature).
- 5. Obtain blood for hematology, biochemistry, serologic tests for HIV and viral hepatitis (B and C), and serological tests for IgE antibodies to *Na*-APR-1 (M74) and *Na*-GST-1.
- 6. Obtain fecal sample for examination for ova and parasites.
- 7. Obtain urine for urine dipstick testing, as well as urine hCG testing in females.
- 8. Counsel females to avoid becoming pregnant during the vaccination phase of the study.

Screening steps 3-8 must be performed within 90 days before the planned enrollment into the study. Should this screening window be exceeded before the first vaccination, screening procedures (not including administration of the informed consent form or comprehension questionnaire) may be repeated to ensure continued eligibility for the study (screening procedures can be repeated a maximum of one time). Screening laboratory tests (other than serologic tests for HIV, viral hepatitis, and antigen specific IgE antibodies) may be repeated up to one time to confirm any abnormalities.

If the fecal exam performed during screening demonstrates infection with an intestinal parasite the individual will be treated with an appropriate medication <u>prior</u> to being enrolled in the study and before any vaccinations. Individuals infected with *Ascaris lumbricoides*, hookworm or *Trichuris trichiura* will be treated with three daily 400 mg doses of albendazole; individuals infected with *S. mansoni* or *Taenia* spp. will be treated with a single 60 mg/kg oral dose of praziquantel; and, individuals infected with *Strongyloides stercoralis* will be treated with three 400 mg daily oral doses of albendazole.

## 7.2 Enrollment/Baseline

Volunteers will not be considered enrolled in the study until they have received their first dose of vaccine. In the event that a volunteer is randomized but not enrolled on the day of first vaccination, they will be replaced with an eligible alternate.

### Study Day 0 (Day of First Vaccination)

- 1. Verify that Informed Consent was obtained.
- 2. Verify that all applicable eligibility criteria have been met.
- 3. Perform abbreviated history (including concomitant medications) and physical exam, focusing on any acute complaints.
- 4. Obtain blood for hematology, biochemistry, anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays, and cellular immunology assays.
- 5. For females, obtain a urine sample for hCG testing. Ensure that test is negative before proceeding; a positive test will exclude the volunteer from the trial.
- 6. Record vital signs (blood pressure, oral temperature, and heart rate).
- 7. Administer the vaccine.
- 8. Observe for at least 1 hour after vaccination to evaluate for immediate adverse reactions. During the 1-hour post-immunization wait period, study staff will discuss signs and symptoms of potential AEs.

## 7.3 Follow-up

#### Study Day 1

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints (i.e., AE data collection).
- 2. Record vital signs.

### Study Day 3 +/- 1

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.

#### Study Day 7 +/- 1

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.
- 3. Obtain blood for anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays and cellular immunology assays.

## Study Day 14 +/- 2

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.
- 3. Obtain blood for hematology, biochemistry, anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays, and cellular immunology assays.

## Study Day 28 +/- 4

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.
- 3. Obtain blood for anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays and cellular immunology assays.

## Study Day 56 +/- 7 (Day of Second Vaccination)

- 1. Perform basic history (including concomitant medications) and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Obtain blood for hematology, biochemistry, anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays, and cellular immunology assays.
- 3. For females, obtain a urine sample for hCG testing. Ensure that test is negative before proceeding; a positive test will exclude the volunteer from further vaccinations.
- 4. Record vital signs.
- 5. Administer the vaccine.
- 6. Observe for at least 1 hour after vaccination to evaluate for immediate adverse reactions.

#### Study Day 57 (1 day after Second Vaccination)

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.

#### Study Day 59 (3 +/- 1 days after Second Vaccination)

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.

## Study Day 63 (7 +/- 1 days after Second Vaccination)

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.
- 3. Obtain blood for anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays and cellular immunology assays.

#### Study Day 70 (14 +/- 2 days after Second Vaccination)

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.
- 3. Obtain blood for hematology, biochemistry, anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays, and cellular immunology assays.

## Study Day 84 (28 +/- 4 days after Second Vaccination)

- 1. Perform basic history and physical exam, emphasizing examination of any complaints.
- 2. Record vital signs.
- 3. Obtain blood for anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays and cellular assays.

## Study Day 112 +/- 14 (Day of Third Vaccination)

- 1. Perform basic history (including concomitant medications) and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Obtain blood for hematology, biochemistry, anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays, and cellular immunology assays.
- 3. For females, obtain a urine sample for hCG testing. Ensure that test is negative before proceeding; a positive test will exclude the volunteer from further vaccinations.
- 4. Record vital signs.
- 5. Administer the vaccine.
- 6. Observe for at least 1 hour after vaccination to evaluate for immediate adverse reactions.

## Study Day 113 (1 day after Third Vaccination)

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.

## Study Day 115 (3 +/- 1 days after Third Vaccination)

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.

### Study Day 119 (7 +/- 1 days after Third Vaccination)

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.
- 3. Obtain blood for anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays and cellular immunology assays.

## Study Day 126 (14 +/- 2 days after Third Vaccination)

- 1. Perform basic history and physical exam (including injection site), emphasizing examination of any acute complaints.
- 2. Record vital signs.
- 3. Obtain blood for hematology, biochemistry, anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays, and cellular immunology assays.

#### Study Day 140 (28 +/-4 days after Third Vaccination)

- 1. Perform basic history and physical exam, emphasizing examination of any acute complaints.
- 2. Obtain blood for anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays and cellular immunology assays.
- 3. Obtain stool for examination for ova and parasites.

## Study Day 200 (3 months +/-14 days after Third Vaccination)

- 1. Perform basic history and physical exam, emphasizing examination of any acute complaints.
- 2. Obtain blood for anti-Na-GST-1 and anti-Na-APR-1 (M74) antibody assays, and cellular immunology assays.

## Study Day 290 (6 months +/-14 days after Third Vaccination)

1. Perform basic history and physical exam, emphasizing examination of any acute complaints.

2. Obtain blood for anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays and cellular immunology assays.

## 7.4 Final Study Visit

Study Day 380 (9 months +/-21 days after Third Vaccination)

- 1. Perform basic history and physical exam, emphasizing examination of any acute complaints.
- 2. Obtain blood for anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) antibody assays and cellular immunology assays.
- 3. Obtain stool for examination for ova and parasites.

## 7.5 Early Termination Visit

The following activities will be performed at the early termination visit for subjects who withdraw, or are withdrawn or terminated from the study:

- Obtain interim medical history by interview of subjects and note any changes since the previous visit.
- All concomitant medications will be recorded on the appropriate data collection form (if within 28 days of subject's last vaccination received in the study).
- Information regarding adverse events/Serious Adverse Events will be assessed and recorded on the appropriate data collection form (adverse events will be limited to new-onset chronic medical conditions and SAEs if after 28 days after the third study vaccination).
- A targeted physical examination may be performed by a study clinician licensed to make medical diagnoses and listed on the Form FDA 1572 as the Principal Investigator or co-investigator, if indicated based on review of interim medical history.
- Approximately 10 mL of venous blood may be collected for safety labs and performed by the local clinical laboratory (if prior to Visit 14 and if not recently obtained per study schedule).
- Approximately 40 mL of venous blood may be collected for antibody and cellular assays (if prior to Visit 14 and if not recently obtained).

## 7.6 Unscheduled Visit

Unscheduled visits may occur at any time during the study. Any of the following activities may be performed:

- Review concomitant medications (if prior to 28 days after a study vaccination).
- Review adverse events (if prior to 28 days after a study vaccination).

- Review serious adverse events and new-onset chronic medical conditions
- Obtain medical history by interview of subjects and note any changes since the previous visit (if indicated).
- A targeted physical examination may be performed by a study clinician, if indicated based on review of medical history.
- Examine study vaccination site (if within 14 days after a study vaccination).
- Approximately 10 mL of venous blood will be collected for safety labs and performed by the study clinical laboratory (if indicated).

## 8 STUDY PROCEDURES/EVALUATIONS

### 8.1 Clinical Evaluations

Subjects will be monitored for local and systemic adverse events during specific protocoldefined post-vaccination periods. As with other aluminum hydroxide-adsorbed vaccines, hypersensitivity reactions would be expected to occur within the first 24 hours after receipt of either of the two vaccines, and other severe local or systemic reactions within 72 hours of vaccination. Subjects will therefore be observed for immediate reactions following each vaccination for at least 1 hour, and will have a clinical assessment either in their home or at the study clinic on Days 1, 3, 7, 14 and 28 following each vaccination. If required, transportation to and from the clinical will be provided. A study clinician will also stay in or near Americaninhas for the duration of the trial and will be available to study subjects at all times. Should a subject call on a study clinician to report an adverse event (AE), it will be fully documented in their study chart, and discussed with the Principal Investigator.

All AEs will be graded for severity and relationship to study vaccine, captured on the appropriate case report form (CRF), and followed to resolution. All Serious Adverse Events (SAEs) will be reviewed by a study physician, recorded on the appropriate SAE form, reported according to applicable regulations and guidelines, and followed through to resolution or stabilization by a study physician. Special attention will also be paid to monitoring for the occurrence of Adverse Events of Special Interest (AESIs), which include inflammatory and autoimmune disorders that may potentially be related to the use of an immunostimulatory adjuvant (although none have been associated with the use of GLA-AF, to date).

A DMID Medical Monitor and a local independent medical monitor will be appointed and a Safety Monitoring Committee (SMC) formed to monitor subject safety and to advise the Principal Investigator and co-investigators on trial-related medical questions or problems. The SMC will periodically review data on safety and enrollment, and will review cumulative safety data for evidence of study related AEs, adherence to the protocol, and factors that may affect outcome or study data such as protocol violations and losses to follow up.

## 8.2 Laboratory Evaluations

## **8.2.1 Clinical Laboratory Evaluations**

Using standard techniques, the following tests will be performed at the accredited Carlos Chagas clinical laboratory in Governador Valadares, Minas Gerais, Brazil. One or more of the laboratory parameters may be repeated at any time during the study as determined by the PI, if indicated by an AE. A clinically significant abnormal value should be repeated within 14 days if possible and followed up as clinically relevant.

- 1. Complete blood count plus white blood cell differential (WBC, absolute neutrophil count [ANC], hemoglobin concentration and platelet count)
- 2. Serum creatinine
- 3. Alanine aminotransferase (ALT)
- 4. Serum glucose (random)
- 5. HBsAg ELISA
- 6. HCV antibody assay
- 7. HIV ELISA

Urine hCG testing will be performed using urine pregnancy test kits that have been approved by Brazilian and/or US regulatory agencies. Urine dipstick testing will also be performed at the trial sites using an approved product.

## 8.2.2 Special Assays or Procedures

Anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) IgG antibody and B cell assays will be performed at the Clinical Immunology Laboratory of the Department of Microbiology, Immunology, and Tropical Medicine (MITM) of the George Washington University; the Dermatology, Allergy, and Clinical Immunology (DACI) Reference Laboratory of Johns Hopkins University; and the University of California at San Francisco. All cryopreservation of plasma, sera and peripheral blood mononuclear cells (PBMCs), as well as screening for levels of IgE against *Na*-APR-1 (M74) and *Na*-GST-1 will take place at the clinical immunology laboratory of CPqRR in Belo Horizonte, Minas Gerais, Brazil. Cryopreservation of sera, plasma and PBMCs will be in liquid nitrogen.

#### 8.2.2.1 Anti-Na-APR-1 (M74) and Anti-Na-GST-1 Antibody Assays

Antibodies to *Na*-APR-1 (M74) and *Na*-GST-1 will be measured in serum or plasma of study subjects using two different methods for comparison: a) a conventional qualified indirect enzyme-linked immunosorbent assay (ELISA) technique using a Standard Reference Serum; and, b) a custom made ImmunoCAP (Phadia, Inc.) for each antigen (*Na*-GST-1 and *Na*-APR-1 (M74)). Antigen-specific IgG and IgG subclass antibody levels will be measured by ELISA and ImmunoCAP at baseline and at several time-points post-vaccination as outlined in Section 3 and in Appendix B. For the qualified conventional indirect ELISA, 96 microwell plates are coated with purified recombinant *Na*-APR-1 (M74) or *Na*-GST-1, blocked, and incubated with serial dilutions of a positive "standard reference serum" pool to generate a reference curve from which antibody levels of test sera can be interpolated. After washing, a horseradish peroxidase conjugated goat anti-human antibody will be added and incubated with plates, washed again, incubated with a chromogenic substrate, and antibody levels measured on an ELISA plate reader.

Qualified ELISAs (one each for *Na*-GST-1 and *Na*-APR-1 (M74)) will also be used to detect IgE antibodies to each antigen, as screening tests to determine eligibility for study participation. If

during screening for volunteer participation in the study, serum samples with anti-Na-GST-1 IgE results by ELISA are greater than the reactivity limit, they will then be tested by the ImmunoCAP method for confirmation. The ImmunoCAP method is considered to be the gold standard for measuring levels of antigen-specific IgE in serum. The ImmunoCAP tests will be performed at the DACI Reference Laboratory of Johns Hopkins University.

Surface Plasmon Resonance (SPR) will be used to measure the affinity of antibody interactions with both recombinant antigens. SPR determines the immunoreactivity and affinity of antibody responses in numerous contexts as it measures rates of antibody-antigen association and dissociation based on the Law of Mass Action to assess antibody affinity.

## 8.2.2.2 Enzyme Neutralization Assays

In vitro assays have been developed to measure the functional capacity of antibodies induced by vaccination with recombinant Na-GST-1 or Na-APR-1 (M74) to inhibit or neutralize the activity of the native forms of these proteins. Serum samples collected from study subjects will be tested for their neutralizing capacity at several post-vaccination time points. These assays will be performed at the Clinical Immunology Laboratory of the Department of MITM of the George Washington University

## 8.2.2.3 Memory B Cell Measurement

The ELISPOT method will be used to evaluate induction of memory B cells (MBCs) after each vaccination and maintenance of MBCs throughout the vaccination schedule to determine if MBCs act as surrogate markers (biomarkers) for later antibody production.

## 8.2.2.4 Cellular Immunology Assays

Cytokine and chemokine assays will be performed on supernatants from cryopreserved PBMCs collected at various time points in the study, by separating PBMCs from whole blood and culturing cells with media only, the mitogen phytohemagglutinin, the antigens Na-APR-1 (M74) or Na-GST-1, and crude Na-americanus antigens extracts (e.g., adult somatic crude antigen extract). Cytokines (e.g., IL-2, IL-4, IL-5, IL-10, TNF $\alpha$ , and IFN $\gamma$ ) will be quantified using Cytometric Bead Analysis kits of supernatants collected from PBMCs stimulated with Na-APR-1 (M74) or Na-GST-1 antigen for 48 and 72 hours *in vitro*. Chemokines (e.g., RANTES, MIP1a, MCP-1, and IP-10) will be quantified in supernatants using commercially available ELISA kits.

#### 8.2.2.5 Parasitology Assays

Fecal exams will begin with an ether sedimentation assay to determine parasite infection status (positive or negative). Positive samples will undergo Kato Katz fecal thick smear exams to determine infection intensity (eggs per gram of feces).

## 8.2.3 Specimen Preparation, Handling, and Shipping

## 8.2.3.1 Instructions for Specimen Preparation, Handling, and Storage

Instructions for specimen preparation, handling, and storage are included in the protocolspecific Manual of Procedures, as appropriate.

#### 8.2.3.2 Specimen Shipment

Specimen shipment will occur at intervals during the course of the study following all applicable International Air Transport Association (IATA) requirements and according to the specifics for storage temperature and documentation as detailed in protocol-specific SOPs, as appropriate.

Specimens for clinical screening and safety laboratory evaluations will be transported from the Americaninhas site to the local (clinical) laboratory.

Specimens for immune responses will be shipped from the Americaninhas site to CPqRR in Belo Horizonte, and then transported to the George Washington University in Washington, DC, in a blinded manner in batches as they become available.

## 9 ASSESSMENT OF SAFETY

## 9.1 Specification of Safety Parameters

Safety will be assessed by the frequency and severity of:

- 1. Study vaccine-related serious adverse events occurring from the time of the first study vaccination through approximately 12 months after the last study vaccination.
- 2. Solicited Adverse Events reactogenicity events occurring on the day of each study vaccination through 14 days after each study vaccination:
  - a) Injection site reactions including erythema (redness), induration (hardness)/swelling, pain, and tenderness.
  - b) Systemic reactions including fever, feverishness (chills/shivering/sweating), fatigue (tiredness), malaise (general unwell feeling), myalgia (body aches/muscular pain exclusive of the injection site), arthralgia (joint pain exclusive of the injection site), headache, and nausea.
- Clinical safety laboratory adverse events occurring from the time of each study vaccination through approximately 14 days after each set of vaccinations. Parameters to be evaluated include WBC, ANC, hemoglobin concentration, and platelet count; ALT; and, creatinine.
- 4. Unsolicited Adverse Events non-serious adverse events occurring from the time of the each study vaccination through approximately 28 days after each vaccination.
- 5. New-onset chronic medical conditions occurring from the time of the first study vaccination through approximately 9 months after the last study vaccination.
- 6. Adverse Events of Special Interest occurring from the time of the first study vaccination through approximately 9 months after the last study vaccination.

## 9.2 Methods and Timing for Assessing, Recording, and Analyzing Safety Parameters

#### 9.2.1 Adverse Events

An adverse event (AE) includes any noxious, pathological or unintended change in anatomical, physiological or metabolic functions as indicated by physical signs, symptoms and/or laboratory-detected changes occurring in any phase of the clinical study, whether associated with the study vaccine or placebo, and whether or not considered vaccination related. This includes an exacerbation of pre-existing conditions and intercurrent illnesses.

All AEs will be graded for severity and relationship to study vaccine. A study clinician will be readily available for the duration of the trial to assess AEs. Should a subject call on a study clinician to report an AE, it will be fully documented in their study chart, and discussed with the Principal Investigator.

All AEs will be assessed by the investigator using the following protocol-defined grading system, as or described in Tables 2-5:

Grade 1: Mild - No effect on activities of daily living; no medical

intervention/therapy required

Grade 2: **Moderate** - Partial limitation in activities of daily living (can

complete ≥50% of baseline); no or minimal medical

intervention/therapy required

Grade 3: **Severe** - Activities of daily living limited to < 50% of baseline;

medical evaluation/therapy required

All AEs will have their possible relationship to study vaccine assessed using the following terms:

Definite: Clear-cut temporal association, and no other possible cause.

<u>Probable</u>: Clear-cut temporal association and a potential alternative etiology is not

apparent.

Possible: Less clear temporal association; other etiologies also possible.

Unlikely: Temporal association between the AE and the vaccine or the nature of the

event is such that the vaccine is <u>not</u> likely to have had any reasonable association with the observed illness/event (cause and effect relationship

improbable but not impossible).

Not Related: The AE is completely independent of vaccine administration; and/or evidence

exists that the event is definitely related to another etiology.

The degree of certainty with which an AE can be attributed to administration of study vaccine will be determined by how well the event can be understood in terms of one or more of the following:

- 1. The event being temporally related with vaccination or reproduced on re-vaccination.
- 2. A reaction of similar nature having previously been observed with this type of vaccine and/or formulation.
- 3. The event having often been reported in the literature for similar types of vaccines.

## 9.2.2 Reactogenicity

Reactogenicity events are AEs that are known to occur with types of vaccine similar in composition to those being tested in this study. The following Toxicity Grading Scales will be used to grade solicited local (injection site) and systemic (subjective and quantitative) reactions:

Table 2: Assessment of Solicited or Expected Adverse Event Severity

| Adverse Event | Grade | Severity |
|---|---|---|
| Pain at injection site | 1 | Easily tolerated, does not interfere with activity |
| | 2 | Repeated use of non-narcotic pain reliever for > 24 hours or |
| | | interferes with daily activity |
| | 3 | Any use of narcotic pain reliever or prevents daily activity |
| Tenderness at injection site | 1 | Mild discomfort to touch |
| | 2 | Discomfort with movement |
| | 3 | Significant discomfort at rest |
| Erythema at injection site | 1 | 25 mm – 50 mm |
| | 2 | 51 mm – 100 mm |
| | 3 | > 100 mm |
| Induration/swelling at injection | 1 | 25 mm – 50 mm and does not interfere with daily activity |
| site | 2 | 51 mm – 100 mm or interferes with daily activity |
| | 3 | >100 mm or prevents daily activity |
| Fever (oral) | 1 | 38.0°C – 38.4°C |
| | 2 | 38.5°C – 38.9°C |
| | 3 | >39.0°C |
| Headache | 1 | Easily tolerated, does not interfere with daily activity |
| | 2 | Repeated use of non-narcotic pain reliever for >24 hours or |
| | | interferes with daily activity |
| | 3 | Any use of narcotic pain reliever or prevents daily activity |
| Nausea | 1 | Easily tolerated, does not interfere with daily activity |
| | 2 | Interferes with daily activity |
| | 3 | Prevents daily activity |
| Vomiting | 1 | 1-2 episodes in 24 hours and does not interfere with activity |
| | 2 | > 2 episodes in 24 hours or interferes with daily activity |
| | 3 | Prevents daily activity or requires outpatient IV hydration |
| Myalgia | 1 | Easily tolerated, does not interfere with daily activity |
| | 2 | Interferes with daily activity |
| | 3 | Prevents daily activity |
| Arthralgia | 1 | Easily tolerated, does not interfere with activity |
| | 2 | Interferes with daily activity |
| | 3 | Prevents daily activity |
| Urticaria | 1 Requiring no medications | |
| | 2 | Requiring PO or topical treatment, or IV medication or steroids for |
| | | <24 hours |
| | 3 | Requiring IV medication or steroids for >24 hours |
| Mucocutaneous Reaction / | 1 | Erythema; pruritus or localized macular rash |
| Rash | 2 | Diffuse, maculopapular rash, dry desquamation |
| | 3 | Vesiculation or moist desquamation or ulceration |

Table 3: Assessment of Unsolicited Systemic Adverse Event Severity

| Systemic AE | Mild | Moderate | Severe |
|---|---|---|---|
| - Jotoliilo AL | (Grade 1) | (Grade 2) | (Grade 3) |
| Anorexia | Loss of appetite without decreased oral intake lasting greater than 48 hours | Loss of appetite associated with decreased oral intake without significant weight loss | Loss of appetite associated with significant weight loss |
| Diarrhea | 3 loose stools/24 hours | 4-5 loose stools/24 hours | >6 loose stools or requires outpatient IV hydration |
| Constipation | Not Applicable | Persistent constipation requiring regular use of dietary modifications, laxatives, or enemas | Obstipation with manual evacuation indicated |
| Fatigue | No interference w/activity | Some interference w/activity | Significant, prevents daily activity |
| Arthritis | Mild pain with inflammation, erythema or joint swelling – but not interfering with function | Moderate pain with inflammation, erythema or joint swelling – interfering with function, but not with activities of daily living | Severe pain with inflammation, erythema or joint swelling –and interfering with activities of daily living |
| Vasovagal<br>episode<br>(associated with a<br>procedure of any kind) | Present without loss of consciousness | Present with transient loss of consciousness | Not Applicable |
| Vertigo | Causes no or minimal interference with usual daily activities | Causes greater than minimal interference with usual daily activities | Inability to perform daily activities |
| Cough | Transient- no treatment | Persistent cough; treatment responsive | Paroxysmal cough; uncontrolled with treatment |
| Bronchospasm,<br>Acute | Transient; no<br>treatment;<br>70% - 80% FEV <sub>1</sub><br>of peak flow | Requires treatment;<br>normalizes with<br>bronchodilator;<br>FEV <sub>1</sub> 50% - 70%<br>(of peak flow) | No normalization with bronchodilator; FEV <sub>1</sub> 25% - 50% of peak flow; or retractions present |
| Dyspnea | Dyspnea on exertion | Dyspnea with normal activity | Dyspnea at rest |
| Hypersensitivity | Transient flushing or rash | Rash; flushing;<br>urticaria; dyspnea | Symptomatic bronchospasm, with or without urticaria; parenteral medications(s) indicated; allergy-related edema/angioedema; hypotension |

Table 4: Assessment of Basic Body Function Adverse Event Severity

| Vital Signs* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|
| Tachycardia –<br>beats per minute | 101-115 | 116-130 | >130 |
| Bradycardia –<br>beats per minute | 50-54 | 45-49 | <45 |
| Hypertension** (systolic, mm Hg) | 141-150 | 151-155 | >155 |
| Hypertension**<br>(diastolic, mm Hg) | 91-95 | 96-100 | >100 |
| Hypotension** (systolic, mm Hg) | 85-89<br>(and symptomatic) | 80-84<br>(and symptomatic) | <80 |
| Respiratory Rate – breaths per minute | 18-20 | 21-25 | >25 |

<sup>\*</sup>Subject should be at rest for measurement of vital signs

**Table 5: Assessment of Laboratory Adverse Event Severity** 

| HEMATOLOGY | Grade 1<br>(Mild) | Grade 2<br>(Moderate) | Grade 3<br>(Severe) |
|---|---|---|---|
| Hemoglobin | | | |
| Males | 11.0 – 12.0 g/dL | 9.5 – 10.9 g/dL | <9.5 g/dL |
| Females | 10.3 – 11.3 g/dL | 8.5 – 10.2 g/dL | <8.5 g/dL |
| Platelets | 110,000 –<br>130,000/mm <sup>3</sup> | 90,000 –<br>109,999/mm <sup>3</sup> | <90,000/mm <sup>3</sup> |
| WBCs | 10,800 – | 15,001 – | <20,000/mm <sup>3</sup> |
| (increase) | 15,000/mm <sup>3</sup> | 20,000/mm <sup>3</sup> | <b>\20,000</b> /11111 |
| WBCs | 2300 – 3200/mm <sup>3</sup> | 1400 – 2299/mm <sup>3</sup> | <1400/mm <sup>3</sup> |
| (decrease) | 2000 - 0200/11111 | 1400 - 2233/11111 | |
| ANC | 750 – 1000/mm <sup>3</sup> | 500 – 749/mm <sup>3</sup> | <500/mm <sup>3</sup> |
| (decrease) | 700 1000/11111 | 7 45/11111 | 1000/111111 |
| CLINICAL | Grade 1 | Grade 2 | Grade 3 |
| CHEMISTRIES | Orauc 1 | Oldac 2 | Orauc o |
| Serum creatinine | | | |
| Males | 1.5 – 1.7 mg/dL | 1.8 – 2.0 mg/dL | >2.0 mg/dL or |
| | | | requires dialysis |
| Females | 1.5 – 1.7 mg/dL | 1.8 – 2.0 mg/dL | >2.0 mg/dL or |
| | | | requires dialysis |
| ALT | ,,_,, | | |
| Males | 58 – 115 U/L | 116 – 230 U/L | >230 U/L |
| Females | 64 – 128 U/L | 129 – 255 U/L | >255 U/L |

All local (injection-site) reactions occurring within the first 7 days after vaccination will be considered <u>definitely</u> related to vaccination.

<sup>\*\*</sup>With repeat testing at same visit

#### 9.2.3 Serious Adverse Events

An SAE is an AE, whether considered related to a study vaccine or not, meeting one of the following conditions:

- 1. Death during the period of protocol-defined surveillance
- 2. <u>Life threatening</u>: defined as an event that places a subject at immediate risk of death at the time of the event and does not refer to an event that hypothetically might have caused death were it more severe
- 3. <u>Hospitalization</u> during the period of protocol-defined surveillance: defined as at least an overnight stay in the hospital or emergency ward for treatment that would have been inappropriate if administered in the outpatient setting
- 4. Results in a congenital anomaly or birth defect
- 5. Results in a persistent or significant <u>disability or incapacity:</u> defined as a substantial disruption of the study subject's ability to carry out normal life functions
- 6. Any other <u>important medical event</u> that may not result in death, be life threatening, or require hospitalization, may be considered a serious AE when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

## 9.2.4 Procedures to be Followed in the Event of Abnormal Laboratory Test Values or Abnormal Clinical Findings

The Principal Investigator or appropriate co-investigator is responsible for reporting all AE/SAEs that are observed or reported during the study, regardless of the relationship to study products. AE/SAEs, abnormal clinical laboratory test values, or abnormal clinical findings will be documented, reported, and followed appropriately.

## 9.3 Reporting Procedures

#### 9.3.1 Serious Adverse Events

All SAEs will be reviewed by a study physician, recorded on the appropriate SAE form, and followed through to resolution or stabilization by a study physician. All SAEs will be reported by email, telephone or fax within 1 working day of notification of the SAE occurrence to the Principal Investigator, via a scanned PDF version of an SAE form to:

#### Dr. Maria Elena Bottazzi, PhD

Deputy Director,
Sabin Vaccine Institute Product Development Partnership
1102 Bates St., Ste. 550, Houston, TX 77030
832-824-0504, Alt. 713-798-1199, Fax 832-825-0549
Email: bottazzi@bcm.edu

In addition, the Principal Investigator will report all SAEs that are determined to be definitely or probably related to vaccination to the Institutional Review Boards (IRBs) that approved the study

(the IRB of the George Washington University and the local IRB in Brazil) according to the IRB's reporting timelines and using the IRB-specified reporting forms, as the DMID Medical Monitor.

All local and systemic reactions not meeting the criteria for SAE will be captured on the appropriate case report form (CRF). These events will be followed to resolution.

In addition, all SAEs must be submitted within 24 hours of site awareness on an SAE form to the DMID pharmacovigilance contractor, at the following address:

DMID Pharmacovigilance Group
Clinical Research Operations and Management Support (CROMS)
6500 Rock Spring Dr. Suite 650
Bethesda, MD 20814, USA

SAE Hot Line: 1-800-537-9979 (US) or 1-301-897-1709 (outside US)
SAE FAX Phone Number: 1-800-275-7619 (US) or 1-301-897-1710 (outside US)
SAE Email Address: PVG@dmidcroms.com

## 9.3.2 Regulatory Reporting for Studies Conducted Under DMID-Sponsored IND

Not Applicable

## 9.3.3 Regulatory Reporting for Studies Not Conducted Under DMID-Sponsored IND

Following notification from the Principal Investigator, the IND sponsor (Sabin Vaccine Institute) will report events that are both serious and unexpected that are possibly, probably, or definitely related to the vaccine, to the FDA and ANVISA (the Brazilian national regulatory agency) within the required timelines: fatal and life-threatening events within 7 calendar days (by phone, fax, or internet) and all other SAEs in writing within 15 calendar days. All SAEs <u>not</u> listed as possibly, probably, or definitely related will be reported to the FDA and ANVISA at least annually in a summary format.

All Adverse Events of Special Interest (AESIs; see below) will be reported to Sponsor, FDA and ANVISA according to the same procedure as for reporting SAEs, and according to the same timelines as described above.

## 9.3.4 Adverse Events of Special Interest (AESI)

Special attention will be paid to monitoring for the occurrence of certain adverse events termed, "Adverse Events of Special Interest" or AESIs. These include inflammatory and autoimmune disorders that may potentially be related to the use of an immunostimulatory adjuvant (although none have been associated with the use of GLA-AF). The occurrence of the following AESI's will be closely monitored:

- Neuroinflammatory disorders (optic neuritis, multiple sclerosis, demyelinating disease, transverse myelitis, Guillain-Barre syndrome, myasthenia gravis, encephalitis, neuritis, Bell's palsy)
- Musculoskeletal disorders (systemic lupus erythematosus, cutaneous lupus, Sjogren's syndrome, scleroderma, dermatomyositis, polymyositis, rheumatoid arthritis, juvenile rheumatoid arthritis, polymyalgia, rheumatica, reactive arthritis, psoriatic arthropathy, ankylosing spondylitis, spondylarthropathy)
- Gastrointestinal disorders (Crohn's disease, ulcerative colitis, celiac disease)
- Metabolic diseases (autoimmune thyroiditis, Grave's or Basedow's disease, Hashimoto thyroiditis, insulin-dependent diabetes mellitus, Addison's disease)
- Skin disorders (psoriasis, vitiligo, Raynaud's phenomenon, erythema nodosum, autoimmune bullous skin diseases)
- Others (autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura, antiphospholipid syndrome, temporal arteritis, Behcet's syndrome, pernicious anemia, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune glomerulonephritis, autoimmune uveitis, autoimmune cardiomyopathy, sarcoidosis, Stevens-Johnson syndrome).
- Vasculitides

## 9.3.5 Medically-Attended Adverse Events (MAAEs)

Special attention will be paid to recording medically-attended adverse events, which are defined as any clinical symptom or diagnosis (including local symptoms at the injection site or systemic symptoms) for which medical evaluation and/or care is sought from a qualified healthcare professional, outside of a regularly scheduled study visit. Note that MAAEs are <u>not</u> the same as SAEs. Whether or not an AE is an MAAE will be recorded on the appropriate Case Report Form.

#### 9.3.6 Reporting of Pregnancy

Pregnancies occurring in study subjects will be reported on the study-specific Pregnancy Report form. No further study vaccinations will be administered to pregnant subjects, but with the subject's permission all study mandated blood samples will be obtained and the subject will continue in follow-up for safety events. Efforts will be made to follow all pregnancies reported during the course of the study to pregnancy outcome pending the subject's permission.

## 9.4 Type and Duration of Follow-up of Subjects after Adverse Events

AEs will be recorded if they start from the time of the first study vaccination (Day 0) up to 28 days after each dose of study product. AEs limited to new-onset chronic medical conditions will be followed through approximately 9 months after the third study vaccination (Day 380).

## 9.5 Halting Rules

If a dose of study vaccine is considered significantly reactogenic (see below and Section 9.2.2), dose escalation and/or additional vaccinations will be suspended <u>until reviewed by the SMC, Independent Safety Monitor, DMID Medical Monitor, and IND sponsor (SVI)</u>. Any recommendation of the Independent Safety Monitor, DMID Medical Monitor, and SMC to resume or suspend further injections (either for an individual subject, an entire Group, or the full study) will be communicated in writing to the sponsor and Principal Investigator. All communications from the SMC will subsequently be forwarded by the investigators to the IRBs.

The following criteria will be used to define significant reactogenicity:

- One or more participants experience a protocol defined SAE that is determined to be possibly, probably, or definitely related to a study vaccine, **OR**,
- One or more participants experience a protocol defined AESI that is determined to be possibly, probably, or definitely related to a study vaccine, **OR**,
- One or more participants experience a protocol defined Grade 3 hypersensitivity reaction that is possibly, probably or definitely related to a study vaccine, **OR**,
- Two or more participants experience a protocol defined Grade 2 hypersensitivity reaction that is probably or definitely related to a study vaccine, **OR**,
- One or more participants in a single Group (i.e., Group 1, Group 2, etc.) experience the same objective physical finding or laboratory abnormality of Grade 3 or higher (with the exception of isolated Grade 3 erythema or swelling), that is determined to be probably or definitely related to a study vaccine, OR,
- Two or more participants in a single Group experience the same Grade 2 or higher safety laboratory abnormality or Grade 3 clinical AE that is possibly, probably or definitely related to a study vaccine.

The study will be double-blinded until all study subjects have completed their Day 140 visit, after which the Sponsor and investigators will be unblinded. During the double-blinded part of the study, a study subject's randomization code may be unblinded only for safety purposes. This is unlikely to occur, since once a vaccine is administered, knowing which vaccine was given is unlikely to influence the medical management of an AE. This procedure is therefore exceptional and any decision to unblind will be discussed with the sponsor, the Principal Investigator, the Independent Safety Monitor, and the SMC. If deemed necessary for urgent safety reasons, the Independent Safety Monitor, in consultation with the SMC (if possible in a timely manner), may unblind a specific subject without revealing the study blind to the investigators or the Sponsor. Any unblinding will be thoroughly documented. It is to be emphasized that the Independent Safety Monitor may put the study on hold at any time and discuss with the SMC. In the event that the investigators come to know the study code prior to final unblinding, the Principal Investigator must notify the Sponsor immediately. The reasons will be documented by the Principal Investigator and added to the study file.

The decision to completely unblind the study prior to Day 140 or permanently stop the study prior to Day 380 will take the form of a formal recommendation by the SMC to the study Sponsor. The Principal Investigator must then notify the IRBs of this decision.

## 9.6 Safety Oversight

## 9.6.1 Independent Safety Monitor (ISM)

An independent Safety Monitor will be appointed for oversight of subject safety in this trial. The ISM will be a local, qualified physician who will be available to advise the investigators on trial-related medical questions or problems. The ISM will work with the DMID Medical Monitor to ensure adequacy of adverse event monitoring and reporting. Should the ISM not be available, he/she will recommend an alternative to serve as a substitute ISM.

The ISM primary responsibility will be to monitor subject safety. The Principal Investigator is responsible for ensuring that the ISM is aware of any new safety information that becomes available during the course of the trial.

## 9.6.2 Safety Monitoring Committee (SMC)

At <u>least</u> three individuals will be selected to serve as the study Safety Monitoring Committee (SMC) to advise the Sponsor and the study investigators on the trial. All SMC members will be independent from the Sponsor and study site. The SMC's primary responsibility will be to monitor subject safety. The Principal Investigator is responsible for ensuring that the SMC is aware of all new safety information. The SMC will periodically review data on safety and enrollment, and will review cumulative safety data for evidence of study related AEs, adherence to the protocol, and factors that may affect outcome or study data such as protocol violations and losses to follow up.

Cumulative safety data reports from the trial will be submitted to the SMC <u>before</u> beginning vaccinations in Group 3 and Group 5 of the study. These safety data reports will include data from at least the first 14 days after first vaccination of all subjects in the prior Group. After the third and final vaccination has been administered to all cohorts, additional safety and immunology results and reports will be submitted to the SMC as they become available.

Conference calls between the investigators and the SMC will be scheduled at least one week prior to beginning vaccinations in Group 3 and Group 5 of the study. If no criteria for halting the study are met (see Section 9.5 above) vaccinations will proceed with approval from the SMC.

Written approval (via fax or email) to proceed to vaccinating Group 3 and Group 5 <u>must</u> be obtained from the SMC prior to vaccine administration. Both the SMC and ISM will have access to the randomization code, as they may wish to review the data in an unblinded fashion should significant safety questions arise prior to the final unblinding of the study.

It is the Principal Investigator's (or designated agent) responsibility to ensure that the SMC reviews the current safety data (grouped by dose cohort), study protocol, and any other requested documents at its meetings. Occurrence of an SAE will be reported to the SMC at the same time that it is reported to the IRBs. Additionally, any new information that may adversely affect the safety of the subjects or the conduct of the study will be submitted to the SMC as it becomes available.

## 10 CLINICAL MONITORING

## 10.1 Site Monitoring Plan

The Sponsor (or its designee) will monitor all aspects of the study, with respect to current Good Clinical Practices, and for compliance with applicable government regulations. Prior to the start of the study, the Principal Investigator will be informed of the frequency of monitoring visits and will be given reasonable notification prior to each visit. The objectives of a monitoring visit will be to verify the prompt reporting of SAEs, to check the availability of the signed Informed Consent for enrolled study subjects, to compare CRFs and spreadsheets with source data for completeness and accuracy, to verify compliance with the clinical protocol, and to check investigational product accountability. During the monitoring visit, the Principal Investigator (and/or designee) and other study personnel should be available to discuss the study. Study documents must be available for review throughout the course of the study.

STATISTICAL CONSIDERATIONS

## 11.1 Study Hypotheses

11

This study is not designed to statistically test a specific hypothesis. Rather, it is intended to assess the safety, reactogenicity, and immunogenicity of two novel vaccines being coadministered to humans for the first time. The chosen sample size principally facilitates the assessment of <u>safety</u>, as discussed in Section 11.2, *Sample Size Considerations*. Given that, this study will <u>explore</u>, primarily by using descriptive statistics, to assess the following hypotheses:

- Co-administration of the Na-APR-1 (M74)/Alhydrogel<sup>®</sup> and Na-GST-1/Alhydrogel<sup>®</sup> vaccines will not increase the reactogenicity or safety risk above that of either administered alone.
- 2. Co-administration of the *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> and *Na*-GST-1/Alhydrogel<sup>®</sup> vaccines will not decrease the functional activity of induced IgG antibodies to either antigen compared to when either is administered alone.
- 3. Co-administration of the *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> and *Na*-GST-1/Alhydrogel<sup>®</sup> vaccines will not decrease the IgG antibody response to either antigen compared to when either is administered alone.
- 4. Co-administration of the *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> and *Na*-GST-1/Alhydrogel<sup>®</sup> vaccines will not decrease the avidity of induced IgG antibodies to either antigen compared to when either is administered alone.
- 5. Co-administration of the *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> and *Na*-GST-1/Alhydrogel<sup>®</sup> vaccines will not decrease the induction of specific MBCs to either antigen compared to when either is administered alone.

## 11.2 Sample Size Considerations

This Phase 1 trial is not powered to detect statistically significant differences between groups. Even though comparative statistics for the safety variables will be computed, the study will have low power to detect anything other than very large differences in the incidence of local injection site and systemic side effects between the vaccination groups. This is done weighing the need to detect any possible untoward reactions against the need to limit the number of volunteers involved for safety purposes. The sample size of 60 for this study is within the range commonly used in Phase 1 trials for the initial assessment of the safety, tolerance and immunogenicity of investigational vaccines.

The primary objective of the study is to estimate the frequency of vaccine-related adverse events. Therefore, rather than providing a statistical power calculation for a specific hypothesis, we illustrate below the probability of observing one or more events, such as an adverse event of a particular type, for a single vaccine dose (N=20), formulation (N=30), or for all participants (N=60) under different assumptions of the true rate at which such events occur in the population.

| | Probability of Observing 1 or More Events | | |
|---|---|---|---|
| | N=20 | N=30 | N=60 |
| "True" (but unknown) Probability of an Event | | | |
| 0.5% | 9.54% | 13.96% | 25.97% |
| 1.0% | 18.21% | 26.03% | 45.28% |
| 3.0% | 45.62% | 59.90% | 83.92% |
| 5.0% | 64.15% | 78.54% | 95.39% |
| 10.0% | 87.84% | 95.76% | 99.82% |

As illustrated in the table above, the study will have high probability (>= 80%) of detecting events that are commonly occurring in the population. For example, with a sample of 20 participants (which is equivalent to the size of each dose group of *Na*-APR-1 (M74) in this study), there is an 87.84% probability of observing 1 or more events when the events occur at a rate of 10.0% in the population. As the sample size increases, the study is able to detect events that occur at lower rates. For example, using a sample size of 30 participants (which is equivalent to the number of participants assigned to vaccine co-administration in this study vs. *Na*-APR-1 (M74) alone), there is a 78.54% probability of observing 1 or more events that occur at a rate of 5% in the population. Using a sample of size 60 (equivalent to the entire study population) there is an 83.92% probability of observing 1 or more events that occur at a rate of 3% in the population. Detection of rare events—those that occur at a rate of 1% or less in the population--is not likely in this study.

## 11.3 Planned Interim Analyses

## 11.3.1 Safety Review

Descriptive and hypothesis-testing approaches will be used to estimate AE rates and to compare these rates in the difference doses and formulations of *Na*-APR-1 (M74) alone or coadministered with *Na*-GST-1. Estimates will be presented with their 95% confidence intervals. Formal statistical tests, as outlined below, will be used to compare doses. No formal adjustments for multiple comparisons will be made. Statistical tests will use a two-sided significance level of 5%.

The proportion of subjects with at least one injection site AE will be compared by vaccine allocation (e.g., *Na*-APR-1 (M74) *vs. Na*-APR-1 (M74) co-administered with *Na*-GST-1), by *Na*-APR-1 (M74) dose, and by GLA-AF dose.

Laboratory results (hematological and clinical chemistry) will be examined for trends over time and any clinically significant values for individuals will be reported.

## 11.3.2 Immunogenicity Review

The proportion of subjects with detectable anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) responses, and the duration of responses, will be summarized as descriptive measures. Geometric mean antibody responses will be compared between Groups with comparisons made by analysis of variance (ANOVA) tests and pair-wise comparisons by contrasts. Antibody responses will be measured at Days 0, 7, 14, 28, 56, 63, 70, 84, 112, 119, and 126 for interim analysis, with Days 140, 200, 290, and 380 added for final analysis.

To exploit the multiple measures of antibody within each subject, a longitudinal model may be built (if possible) to describe the antibody responses over time. The models will explore if there are any differences between those administered *Na*-APR-1 (M74)/Alhydrogel<sup>®</sup> alone and those co-administered *Na*-GST-1/Alhydrogel<sup>®</sup>.

Summary statistics will be used to present exploratory study results of the cellular immune responses to *Na*-GST-1 and *Na*-APR-1 (M74) before and after immunization. To assess the changes in lymphocyte proliferative responses and cytokine/chemokine profiles over time, a generalized estimating equations model with robust standard errors will be constructed. When necessary, data reduction approaches will be used.

## 11.4 Final Analysis Plan

The purpose of this trial is to estimate AE rates and patterns of immune response as well as to compare these rates and patterns between the investigational vaccines, when they are administered separately or when they are co-administered.

This section briefly describes the statistical methods to be used; a detailed analytical plan will fully describe the methods. The analytical plan will discuss the planned approaches to missing data. Deviations from the original analytical plan will be thoroughly documented and reported to the Sponsor.

Descriptive and hypothesis-testing approaches will be used to meet the protocol objectives as stated in **Section 3**. Estimates will be presented with their 95% confidence intervals. Formal statistical tests, as outlined below, will be used to compare doses. Statistical tests will use a two-sided significance level of 5%.

Note: For the analyses described below, historical safety data from a Phase 1 clinical trial conducted at the same study site and in the same subject population (study SVI-10-01, see **Section 2.1.6** above for a description of this trial) will be used to obtain a comparison of *Na*-GST-1/Alhydrogel. As well, stored serum and cell specimens from those study participants will be used in the immunological assays to obtain data on subjects administered *Na*-GST-1/Alhydrogel without co-administered *Na*-APR-1 (M74). These specimens from SVI-10-01 will be assayed at the same time as those newly collected from the study described in this protocol.
<u>Primary Objective</u>: To evaluate the safety and reactogenicity of three different dose concentrations of *Na*-APR-1 (M74) adjuvanted with Alhydrogel<sup>®</sup> or Alhydrogel<sup>®</sup> plus GLA-AF and administered either with or without *Na*-GST-1, in healthy Brazilian adults.

AEs will be coded according to Medical Dictionary of Regulatory Activities (MedDRA<sup>TM</sup>) preferred terms. The frequency, severity, and relationship of AEs per each vaccine formulation and dose cohort of *Na*-APR-1 (M74) and co-administration status with *Na*-GST-1 will be presented in tabular form using the MedDRA<sup>TM</sup> coded term and organized by MedDRA<sup>TM</sup> System, Organ, and Class (SOC) designations.

- The frequency of immediate, systemic, and local injection site AEs will be summarized by SOC and preferred term.
- Line listings of clinical and laboratory AEs classified as immediate (within the first 60 minutes), systemic, and local will be displayed in tables stratified by dose cohort and formulation of *Na*-APR-1 (M74) and formulation (i.e., no GLA-AF or 5 µg GLA-AF).
- AEs will be summarized by severity and relationship to vaccine formulation by individuals and dose of *Na*-GST-1, *Na*-APR-1 (M74), and GLA-AF.
- The frequency of vaccine-related SAEs will be tallied as well as summarized by body system, by vaccine formulation and dose cohort.

### Primary Outcome Measures:

The following summary parameters will be evaluated for each dose and formulation of *Na*-APR-1 (M74) alone or co-administered with *Na*-GST-1:

- 1. Frequency of solicited injection site and systemic reactogenicity, graded by severity, on the day of each study vaccination through 14 days after each study vaccination.
- 2. Frequency of study vaccine-related serious adverse events from the time of the first study vaccination through approximately 9 months after the last study vaccination.
- 3. Frequency of clinical safety laboratory adverse events.
- 4. Frequency of unsolicited adverse events, graded by severity, from the time of each study vaccination through approximately 1 month after each study vaccination.
- 5. Frequency of new-onset chronic medical conditions through approximately 9 months after the third study vaccination.
- 6. Frequency of Adverse Events of Special Interest through approximately 9 months after the third study vaccination.

### Analysis Plan:

The proportion of participants with at least one injection site AE will be compared by *Na*-APR-1 (M74) vaccine formulation and dose cohort and co-administration status with *Na*-GST-1. We will test the null hypotheses that the type and number of adverse events is the same across all groups by Fisher's exact test.

Laboratory results (hematological and clinical chemistry) will be examined for trends over time and any clinically significant values for individuals will be reported.

<u>Secondary Objective</u>: To assess the impact of co-administering *Na*-APR-1 (M74) and *Na*-GST-1 on antibody production by measuring the antibody levels to each antigen on study Day 126.

### Secondary Outcome Measures:

The following parameters will be evaluated for each dose and formulation of *Na*-APR-1 (M74) alone or co-administered with *Na*-GST-1:

- 1. The IgG level by an indirect enzyme-linked immunosorbent assay (ELISA) on approximately Day 126.
- 2. The IgG level by ImmunoCAP on approximately Day 126.

## Analysis Plan:

- a. The proportion of participants with detectable anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) responses will be summarized as a descriptive measure.
- b. IgG levels will be displayed graphically by study group using notched box plots.
- c. Geometric mean antibody responses will be compared between vaccine formulation and dose groups. Comparisons between groups will be made by a one-way analysis of variance (ANOVA) with pair-wise comparisons between groups made by contrasts.
- d. Geometric mean antibody responses for each antigen will be compared using a regression model with main effects for the doses of Na-APR-1 (10, 30 or 100μg), GLA-AF (0 or 5 μg), and Na-GST-1 (0, 100μg).
- e. For antigen-specific log IgG levels, a three-way ANOVA will be conducted, with *Na*-GST-1, *Na*-APR (M74) and GLA-AF doses as factors.
- f. Pair-wise comparisons across all combinations of Na-APR-1 (M74) doses, GLA-AF doses (i.e., 0 or 5  $\mu$ g), and Na-GST-1 co-administration status will be assessed using Tukey's HSD.

<u>Tertiary Objective 1</u>: To assess the impact of co-administration of *Na*-GST-1 on the duration of the antibody responses to *Na*-APR-1 (M74), and vice versa.

Tertiary Outcome Measure 1: The IgG antibody response, by an indirect enzyme-linked immunosorbent assay (ELISA) at approximately 7, 14, and 28 days after each vaccination, and approximately 3, 6, and 9 months after the third dose.

Tertiary Outcome Measure 2: The IgG antibody response, by ImmunoCAP at approximately 7, 14, and 28 days after each vaccination, and approximately 3, 6, and 9 months after the third dose.

### Analysis Plan:

- a. The proportion of participants with detectable anti-*Na*-GST-1 and anti-*Na*-APR-1 (M74) responses will be summarized as a descriptive measure.
- b. Antigen-specific IgG levels will be displayed graphically by study group using notched box plots at each time point.

c. Geometric mean antibody responses will be compared between vaccine formulation and dose groups at each time point. Comparisons between groups will be made by a

one-way analysis of variance (ANOVA) with pair-wise comparisons between groups made by contrasts.

d. Percent change in IgG antibody levels from days of vaccination to days 7,14 and 28 will be compared between vaccine formulation and dose groups. Values will be reported with 95% confidence intervals.

- e. Percent change in IgG antibody levels from vaccination day #1 to #2, and from vaccination day #2 to #3 will be compared between vaccine formulation and dose groups to assess the sustainability of the response from trough to trough. Values will be reported with 95% confidence intervals.
- f. Percent change in IgG antibody levels from the peak following the third vaccination, to 3, 6 and 9 months after the third vaccination. Values will be reported with 95% confidence intervals.
- g. Geometric mean antibody responses for each antigen will be compared using a regression model at each time point with main effects for the doses of Na-APR-1 (M74) (10, 30 or 100μg), GLA-AF (0 or 5μg), and Na-GST-1 (0, 100μg)
- h. For antigen-specific log IgG levels, three-way ANOVAs will be conducted, with *Na*-APR-1 (M74) dose, GLA-AF dose, and *Na*-GST-1 co-administration status as factors.
- i. A longitudinal model will be built to describe the IgG levels over time. Using a longitudinal panel model, differences in antibody isotype levels by dose and formulation of *Na*-APR-1 (M74) and *Na*-GST-1 co-administration status will be explored. This will be accomplished using Proc Mixed in SAS 9.3 so the analysis will take account of the correlation between measurements on the same participant.

<u>Tertiary Objective 2</u>: To assess the impact of co-administration of *Na*-GST-1 on the distribution of IgG subclass responses to *Na*-APR-1 (M74) and vice versa.

*Tertiary Outcome Measure 3*: The IgG subclass distribution (IgG1, IgG3, and IgG4) by plate based ImmunoCAP on approximately Day 126.

Tertiary Outcome Measure 4: The IgG subclass distribution by plate based ImmunoCAP each day of vaccination, approximately 28 days later, and approximately 3 and 6 months after the final vaccination.

#### Analysis Plan:

- a. The proportion of subjects with detectable anti-Na-GST-1 and anti-Na-APR-1 (M74) lgG subclass responses will be summarized at each time point as a descriptive measure.
- b. IgG subclass antibody levels will be displayed graphically by study group using notched box plots at each time point.
- c. Geometric mean antibody responses will be compared between vaccine formulation and dose groups. Comparisons between groups will be made by a one-way analysis

- of variance (ANOVA) with pair-wise comparisons between groups made by contrasts.
- d. For antigen-specific IgG subclass (IgG1-IgG4) levels, a three-way ANOVA will be conducted, with *Na*-APR-1 (M74) and GLA-AF doses, and *Na*-GST-1 coadministration status, as factors.
- e. A longitudinal model will be built to describe each of the antibody isotype levels over time for each of IgG1-IgG4. Using a longitudinal panel model, differences in antibody isotype levels by dose and formulation of *Na*-APR-1 (M74) and *Na*-GST-1 co-administration status will be explored. This will be accomplished using Proc Mixed in SAS 9.3 so the analysis will take account of the correlation between measurements on the same participant.

<u>Tertiary Objective 3</u>: To assess the impact of co-administration of *Na*-GST-1 and *Na*-APR-1 (M74) on the functional capacity of vaccine-induced antibodies to neutralize the *in vitro* activity of the native enzymes (*Na*-GST-1 and wild type *Na*-APR-1).

*Tertiary Outcome Measure 5*: The functional capacity of vaccine-induced antibodies to neutralize the *in vitro* activity of the native enzymes.

### Analysis Plan:

- a. Percent inhibition of native enzyme activity will be displayed graphically for the various study groups at each time point.
- b. Three-way ANOVAs with *Na*-APR-1 (M74), *Na*-GST-1, and GLA-AF as factors and percent inhibition as the outcome will be estimated.
- c. A longitudinal model will be built to describe percent inhibition of native enzyme activity over time. Using a longitudinal panel model, differences in percent inhibition by dose and formulation of *Na*-APR-1 (M74) and co-administration with *Na*-GST-1 will be explored. This will be accomplished using Proc Mixed in SAS 9.3, so the analysis will take account of the correlation between measurements on the same participant.

<u>Tertiary Objective 4</u>: To assess the impact of co-administration of *Na*-GST-1 and *Na*-APR-1 (M74) on the affinity of the antibody interactions with both recombinant antigens.

Tertiary Outcome Measure 6: The affinity of the antibody interactions with both recombinant antigens at approximately 7, 14, and 28 days after each vaccination, and 3, 6, and 9 months after the third dose.

### Analysis Plan:

- a. Antibody affinity will be displayed graphically for the various study groups at each time point.
- b. Three-way ANOVAs with *Na*-APR-1 (M74), *Na*-GST-1, and GLA-AF as factors and overall affinity as the outcome will be estimated.

c. A longitudinal model will be built to describe increasing antibody affinity (affinity maturation) over time. Using a longitudinal panel model, differences in affinity maturation by dose and formulation of *Na*-APR-1 (M74) and co-administration with *Na*-GST-1 will be explored. This will be accomplished using Proc Mixed in SAS 9.3, so the analysis will take account of the correlation between measurements on the same participant.

<u>Tertiary Objective 5</u>: To assess the impact of co-administration of *Na*-GST-1 and *Na*-APR-1 (M74) on the production of memory B cells specific for each antigen.

Tertiary Outcome Measure 7: The production of memory B cells specific for each antigen on days of vaccination, approximately 28 days following each vaccination, and 6 and 9 months after the third dose.

### Analysis Plan:

- a. The amount of *Na*-GST-1 and *Na*-APR-1 (M74) specific memory B cells will be expressed as a percentage of total lymphocytes present in the blood.
- b. The percentage of specific memory B cells will be displayed graphically by study group at each time point.
- c. Two separate longitudinal panel analyses will test the null hypothesis that average percentages for each of memory B cells are the same in *Na*-APR-1 (M74) groups with and without co-administration of *Na*-GST-1 over time. This will be accomplished using Proc Mixed in SAS 9.3 so the analysis will take account of the correlation between measurements on the same participant.
- d. Mann-Whitney tests will assess the null hypothesis that cytokine levels are the same in the groups at the primary time point of Day 126, two weeks after final vaccination.

<u>Exploratory Objective</u>: To assess the cellular immune responses to the *Na*-GST-1 and *Na*-APR-1 (M74) antigens following immunization.

The following assays will be performed to assess the cellular immune responses to vaccination with *Na*-APR-1 (M74) +/- *Na*-GST-1:

- a. Lymphocyte proliferative responses to *in vitro* stimulation with *Na*-GST-1 or *Na*-APR-1 (M74).
- b. Cytokine and chemokine production *in vitro* in response to stimulation with *Na*-GST-1 or *Na*-APR-1 (M74).
- c. Changes in *in vivo* PBMC subpopulations as determined by flow cytometry.
- d. A longitudinal panel analysis will test the null hypothesis that cytokine and chemokine levels are the same when *Na*-APR-1 (M74) is administered with and without or *Na*-GST-1 and examine for trends over time.

·

Should the study be terminated early, the investigative team will discuss with the SMC the reason for termination and determine which study questions can be addressed in an unbiased manner with the available data. The available data will be analyzed and interpreted in light of early termination.

12 SOURCE DOCUMENTS AND ACCESS TO SOURCE DATA/DOCUMENTS

Complete source documentation (clinical evaluations and test results) will be collected for every study subject for the duration of the study, with supplementary documents (laboratory test reports, supplementary hospital or medical records, etc.) forming part of the source documentation. Case Report Forms (CRFs) will be used to record study-specific data for enrolled subjects, and study-specific data may be entered directly onto CRFs: in these cases, the documents will be both source and CRF. The Principal Investigator will responsible for the accuracy and completeness of the data reported in the CRFs and the source documents. Data reported in the CRFs that is derived from source documents should be consistent with source documents and the discrepancies should be explained.

# 13 QUALITY CONTROL AND QUALITY ASSURANCE

Following a written Sponsor-accepted site quality management plan, the investigational site is responsible for conducting routine quality assurance and quality control activities to internally monitor study progress and protocol compliance. The PI will provide direct access to all trial-related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities. The PI will ensure all study personnel are appropriately trained and applicable documentation is maintained on site.

Clinical monitors will verify that the clinical trial is conducted and data are generated, documented (recorded), and reported in compliance with the protocol, ICH/GCP guidelines, and the applicable regulatory requirements. Clinical monitoring reports will be submitted to the Sponsor.

The data management vendor will implement quality control procedures beginning with the data entry system and generate data quality control checks that will be run on the database. Any missing data or data anomalies will be communicated to the site(s) for clarification and resolution.

## 14 ETHICS/PROTECTION OF HUMAN SUBJECTS

The study will be conducted according to fundamental ethical principles including: The principle of respect for human dignity and the principles of non-exploitation, non-discrimination and non-instrumentalisation; The principle of individual autonomy (entailing the giving of free and informed consent, and respect for privacy and confidentiality of personal data); The principle of justice (the equitable distribution of burdens and benefits of research); The principle of beneficence and non-maleficence, namely with regard to the improvement and protection of health; and, The principle of proportionality (including that research methods are necessary to the aims pursued and that no alternative more acceptable methods are available).

## 14.1 Ethical Standard

The study will be conducted according to: the Declaration of Helsinki (amended in 2008); CIOMS (Council for International Organizations of Medical Sciences) International Ethical Guidelines for Biomedical Research Involving Human Subjects (2002); International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) (1996) Guideline for good clinical practice E6 (R1); the US Code of Federal Regulations (Protection of Human Subjects [21 CFR 50], Institutional Review Boards [21 CFR 56], and Obligations of Clinical Investigators [21 CFR 312]); and, Brazilian Resolution N° 466/12 (that replaced Resolution N° 196/96) on Research Involving Human Subjects.

### 14.2 Institutional Review Boards

The investigators will be responsible for obtaining full IRB approvals for the study from the local Brazilian IRB (at the Federal University of Minas Gerais) and George Washington University IRBs. Before the start of the study, the appropriate documents (including the protocol, Investigator's Brochures, and informed consent form) will be submitted to the IRBs. The IRBs will be informed by the Investigator of any new information that may adversely affect the safety of the subjects or the conduct of the study, an annual update and/or request for re-approval, and when the study has been completed

### 14.3 Informed Consent Process

The principles of informed consent in the current edition of the Declaration of Helsinki will be implemented and informed consent obtained in accordance with US 21 CFR 50.25 and Brazilian Resolution Nº 466/12 on Research Involving Human Subjects. For SVI-DBL-01 a community meeting will be held to provide volunteers with an overview of the clinical trial and study procedures, and to answer questions in an open forum. This group meeting will be followed by individual informed consent sessions with each interested volunteer. Individual sessions may be on the same day as the community meeting, or scheduled for a later date. During the individual session a member of the study team will read the consent form together with the volunteer, regardless of whether or not the volunteer is illiterate. The study team member will explain why the volunteer is being invited to participate in the study and will clarify all of the volunteer's

questions. Throughout the informed consent process volunteers will be encouraged to ask questions, and if they wish, to discuss the study with family or community members prior to making their decision.

Volunteers agreeing to participate will first provide written informed consent and take a true/false comprehension questionnaire. The questionnaire is administered orally in the case of illiterate volunteers, and for both written and oral questionnaires study staff will use incorrect answers to identify aspects of the study that require clarification and focus on those areas of the informed consent form for further review with the volunteer. All questionnaire questions must be answered correctly, and the informed consent form signed, prior to study screening and enrollment. Volunteers unable to read will place an imprint of their finger in the place of a signature; in addition, an independent witness, who is not a member of the study team, will sign the consent form to attest that the informed consent form was read to the volunteer, the volunteer's questions were answered, and the volunteer answered all comprehension questions correctly. The original signed informed consent form for each volunteer will be maintained as part of that volunteer's study records. A copy of the informed consent form will be provided to every volunteer.

### 14.3.1 Informed Consent/Assent Process (in Case of a Minor)

Not Applicable

# 14.4 Exclusion of Women, Minorities, and Children (Special Populations)

Healthy adults age 18 to 45 meeting all protocol defined inclusion and exclusion criteria will be invited to participate. Females of childbearing potential, unless surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), at least 2 years postmenopausal, or practicing abstinence, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner) until at least one month following the last immunization. Female participants will be counseled by a study clinician or nurse, or referred to the local health center for evaluation and institution of an appropriate contraceptive method.

This clinical trial will enroll healthy, non-pregnant volunteers from the general population of the a study site in the Brazilian state of Minas Gerais located in and around the town of Americaninhas, without regard to gender or racial/ethnic group. That is, no specific racial/ethnic groups will be targeted or excluded from participation in these trials. In addition, both (non-pregnant) women and men will be equally encouraged to participate, and it is expected that roughly equal numbers of each gender will consent to participate in this Phase 1 study, based on the experience of the study team that will conduct the proposed clinical trial and which has enrolled subjects into similar vaccine trials at the same site.

There will not be any research conducted on children under the age of 18 years as part of this trial. Children between the ages of 18-21 years, inclusive, will be eligible to participate in this Phase 1 trial, given that the legal age of consent in Brazil is 18 years.

·

# 14.5 Subject Confidentiality

All study-related information will be stored securely at the study site. All subject information will be stored in locked file cabinets in areas with access limited to study staff. All laboratory specimens, reports, study data collection, and administrative forms will be identified by coded numbers only, to maintain subject confidentiality. All computer entries will also be made using coded number only, and all local databases will be secured with password-protected access systems. Forms, lists, and any other listings that link subject identification numbers to other identifying information will be stored in a separate, locked file in an area with limited access.

Subject study information will not be released without the written permission of the subject, except as necessary for monitoring by the sponsor and/or its designee, the US National Institutes of Health, and the FDA or Brazilian regulatory authorities.

# 14.6 Study Discontinuation

If the trial is discontinued, subjects who sign the informed consent form, and are randomized and vaccinated will continue to be followed for safety assessments. No further study vaccinations will be administered.

# 14.7 Future Use of Stored Specimens

Some of the biological samples collected from study participants may be stored at the local site and some at CPqRR in Belo Horizonte or at the MITM at GWU. Stored samples may be shared with other investigators at other institutions for the purposes of conducting the tests outlined in this study protocol. Stored samples will not be sold or used directly for production of any commercial product. No human genetic tests will be performed on samples. Each sample will be encoded (labeled) only with a unique code and a unique tracking number to protect subject's confidentiality. There are no benefits to subjects in the collection, storage and subsequent research use of samples. Reports about research done with subject's samples will NOT be kept in their health records. Any proposed future research using samples collected from study participants will first be submitted to the applicable IRBs for approval. The IRBs will determine if the study participants must be re-consented for the use of their samples in such research.

DATA HANDLING AND RECORD KEEPING

# 15.1 Data Management Responsibilities

All data collection forms and laboratory reports must be reviewed by the clinical team and data entry personnel, who will ensure that they are accurate and complete. Adverse events must be recorded on the appropriate data collection form, assessed for severity and relationship to vaccination, and reviewed by the Principal Investigator or appropriate co-investigator.

Data collection is the responsibility of the study personnel at the study site under the supervision of the Principal Investigator. During the study, the Principal Investigator must maintain complete and accurate documentation for the study.

The data management vendor for this study will be responsible for data management, quality review, analysis, and reporting of the study data.

# 15.2 Data Capture Methods

CRFs will be used to record study-specific data for enrolled subjects, and study-specific data may be entered directly onto CRFs: in these cases, the documents will be both source and CRF. The Principal Investigator will responsible for the accuracy and completeness of the data reported in the CRFs and the source documents. Data reported in the CRFs that is derived from source documents should be consistent with source documents and the discrepancies should be explained.

# 15.3 Types of Data

15

Data for this study will include clinical, safety, and outcome measures (e.g., clinical laboratory values, reactogenicity, and immunogenicity data).

# 15.4 Timing/Reports

In addition to the study-related documentation required by the regulatory authorities, 4 study reports will be generated. These include 2 interim SMC safety reports, 1 interim safety and immunogenicity study report, and the final study report. The first interim SMC safety report will be completed after the safety data from the Day 14 visits of Group 2 have been compiled, for the purposes of deciding whether it is safe to precede with enrollment into Group 3 of the study. The second interim SMC safety report will be completed after the safety data from the Day 14 visits of Group 4 have been compiled, for the purposes of deciding whether it is safe to precede with enrollment into Group 5 of the study. The interim study report will be compiled after interim safety and primary immunogenicity data (i.e., antigen-specific IgG responses to *Na*-GST-1 and *Na*-APR-1 (M74) as determined by ELISA) from all Day 140 visits is available and the study investigators unblinded. This report will serve as the basis for deciding whether to continue with

·

future Phase 1 testing of the vaccines in children. A final report containing all safety and immunology data will be prepared after trial completion.

# 15.5 Study Records Retention

Trial-related documents will be maintained by the Investigator for a period of 2 years after final marketing approval of the vaccine, or if 2 years have elapsed since the formal discontinuation of clinical development of the product. During the study and while archived at the site all study-related information will be stored securely in locked file cabinets in areas with access limited to study staff. All laboratory specimens, reports, study data collection, and administrative forms will be identified by coded number only, to maintain subject confidentiality. All computer entries will be done using a coded number only, and all local databases will be secured with password-protected access systems. Forms, lists, and any other listings that link subject ID numbers to other identifying information will be stored in a separate, locked file in an area with limited access. Subject study information will not be released without the written permission of the subject, except as necessary for monitoring, and the FDA or Brazilian regulatory authorities.

### 15.6 Protocol Deviations

No modifications to this protocol will be implemented without prior written IRB approval. This does not apply to changes made to reduce discomfort or avert risk to study subjects. Furthermore, in the event of a medical emergency, the investigators shall perform any medical procedures that are deemed medically appropriate. The Principal Investigator must notify the Sponsor and IRBs of all such occurrences. Any change to the protocol will be submitted to the actively participating IRBs as a protocol amendment, and changes not affecting risk to subjects may be expedited, as appropriate.

Any deviation from the IRB approved protocol will be documented, including the date and detailed description of the deviation and all corrective actions taken. For any deviation determined to have potential or known impact on subject safety, an IRB problem report will be generated and submitted to the IRBs according to their guidelines and reporting timelines.

# 16 PUBLICATION POLICY

It is anticipated that results from this study will be published in peer-reviewed journals. If publication is sought, the identity of study subjects or any easily traceable identifiers will not be revealed. Authorship issues will be discussed and agreed upon between the Sponsor and collaborating partners prior to submission for publication. Additionally, the results of the study will be communicated to both study subjects and the community at large.

The Principal Investigator and all partners on this study will make publically available any final research data resulting from the trial, in a timely fashion following closure of the clinical trial (not more than 12 months after the last subject follow-up visit).

## 17 LITERATURE REFERENCES

1. Ashford RW, Craig PS, Oppenheimer SJ. Polyparasitism on the Kenya coast. 1. Prevalence, and association between parasitic infections. Ann Trop Med Parasitol 1992;86:671-679.

- 2. de Silva NR, Brooker S, Hotez PJ, Montresor A, Engels D, Savioli L. Soil-transmitted helminth infections: updating the global picture. Trends Parasitol 2003;19:547-551.
- 3. Hotez PJ, Brooker S, Bethony JM, Bottazzi ME, Loukas A, Xiao S. Hookworm infection. N Engl J Med 2004;351:799-807.
- 4. Stoltzfus RJ, Chwaya HM, Montresor A, Albonico M, Savioli L, Tielsch JM. Malaria, hookworms and recent fever are related to anemia and iron status indicators in 0- to 5-y old Zanzibari children and these relationships change with age. J Nutr 2000;130:1724-1733.
- 5. Stoltzfus RJ, Dreyfuss ML, Chwaya HM, Albonico M. Hookworm control as a strategy to prevent iron deficiency. Nutr Rev 1997;55:223-232.
- 6. Guyatt HL, Brooker S, Peshu N, Shulman CE. Hookworm and anaemia prevalence. Lancet 2000;356:2101.
- 7. Brooker S, Bethony J, Hotez PJ. Human hookworm infection in the 21st century. Adv Parasitol 2004;58:197-288.
- 8. Brooker S, Peshu N, Warn PA, Mosobo M, Guyatt HL, Marsh K, Snow RW. The epidemiology of hookworm infection and its contribution to anaemia among pre-school children on the Kenyan coast. Trans R Soc Trop Med Hyg 1999;93:240-246.
- 9. Bundy DA, Chan MS, Savioli L. Hookworm infection in pregnancy. Trans R Soc Trop Med Hyg 1995;89:521-522.
- 10. Stoltzfus RJ, Chwaya HM, Tielsch JM, Schulze KJ, Albonico M, Savioli L. Epidemiology of iron deficiency anemia in Zanzibari schoolchildren: the importance of hookworms. Am J Clin Nutr 1997;65:153-159.
- 11. Guyatt HL, Brooker S, Kihamia CM, Hall A, Bundy DA. Evaluation of efficacy of school-based anthelmintic treatments against anaemia in children in the United Republic of Tanzania. Bull World Health Organ 2001;79:695-703.
- 12. Sakti H, Nokes C, Hertanto WS, Hendratno S, Hall A, Bundy DA, Satoto. Evidence for an association between hookworm infection and cognitive function in Indonesian school children. Trop Med Int Health 1999;4:322-334.
- 13. Jardim-Botelho A, Raff S, Rodrigues Rde A, Hoffman HJ, Diemert DJ, Correa-Oliveira R, Bethony JM, et al. Hookworm, Ascaris lumbricoides infection and polyparasitism associated with poor cognitive performance in Brazilian schoolchildren. Trop Med Int Health 2008;13:994-1004.
- 14. Bundy DA, Medley GF. Immuno-epidemiology of human geohelminthiasis: ecological and immunological determinants of worm burden. Parasitology 1992;104 Suppl:S105-119.
- 15. Bethony J, Chen J, Lin S, Xiao S, Zhan B, Li S, Xue H, et al. Emerging patterns of hookworm infection: influence of aging on the intensity of Necator infection in Hainan Province, People's Republic of China. Clin Infect Dis 2002;35:1336-1344.
- 16. Sampathkumar V, Rajaratnam A. Prevalence of anaemia and hookworm infestation among adolescent girls in one rural block of TamilNadu. Indian J Matern Child Health 1997;8:73-75.
- 17. Utzinger J, Keiser J. Schistosomiasis and soil-transmitted helminthiasis: common drugs for treatment and control. Expert Opin Pharmacother 2004;5:263-285.

- 18. Bennett A, Guyatt H. Reducing intestinal nematode infection: efficacy of albendazole and mebendazole. Parasitol Today 2000;16:71-74.
- 19. Horton J. Albendazole: a review of anthelmintic efficacy and safety in humans. Parasitology 2000;121 Suppl:S113-132.
- 20. Keiser J, Utzinger J. Efficacy of current drugs against soil-transmitted helminth infections: systematic review and meta-analysis. JAMA 2008;299:1937-1948.
- 21. Hotez PJ, Zhan B, Bethony JM, Loukas A, Williamson A, Goud GN, Hawdon JM, et al. Progress in the development of a recombinant vaccine for human hookworm disease: the Human Hookworm Vaccine Initiative. Int J Parasitol 2003;33:1245-1258.
- 22. Diemert DJ, Bethony JM, Hotez PJ. Hookworm vaccines. Clin Infect Dis 2008;46:282-288.
- 23. Pullan RL, Bethony JM, Geiger SM, Cundill B, Correa-Oliveira R, Quinnell RJ, Brooker S. Human helminth co-infection: analysis of spatial patterns and risk factors in a Brazilian community. PLoS Negl Trop Dis 2008;2:e352.
- 24. Bethony JM, Simon G, Diemert DJ, Parenti D, Desrosiers A, Schuck S, Fujiwara R, et al. Randomized, placebo-controlled, double-blind trial of the Na-ASP-2 hookworm vaccine in unexposed adults. Vaccine 2008;26:2408-2417.
- 25. Diemert DJ, Pinto AG, Freire J, Jariwala A, Santiago H, Hamilton RG, Periago MV, et al. Generalized urticaria induced by the Na-ASP-2 hookworm vaccine: implications for the development of vaccines against helminths. J Allergy Clin Immunol 2012;130:169-176 e166.
- 26. Ranjit N, Zhan B, Hamilton B, Stenzel D, Lowther J, Pearson M, Gorman J, et al. Proteolytic degradation of hemoglobin in the intestine of the human hookworm Necator americanus. J Infect Dis 2009;199:904-912.
- 27. Williamson AL, Brindley PJ, Abbenante G, Prociv P, Berry C, Girdwood K, Pritchard DI, et al. Cleavage of hemoglobin by hookworm cathepsin D aspartic proteases and its potential contribution to host specificity. FASEB J 2002;16:1458-1460.
- 28. Williamson AL, Brindley PJ, Abbenante G, Datu BJ, Prociv P, Berry C, Girdwood K, et al. Hookworm aspartic protease, Na-APR-2, cleaves human hemoglobin and serum proteins in a host-specific fashion. J Infect Dis 2003;187:484-494.
- 29. Williamson AL, Lecchi P, Turk BE, Choe Y, Hotez PJ, McKerrow JH, Cantley LC, et al. A multi-enzyme cascade of hemoglobin proteolysis in the intestine of blood-feeding hookworms. J Biol Chem 2004;279:35950-35957.
- 30. Loukas A, Bethony JM, Mendez S, Fujiwara RT, Goud GN, Ranjit N, Zhan B, et al. Vaccination with recombinant aspartic hemoglobinase reduces parasite load and blood loss after hookworm infection in dogs. PLoS Med 2005;2:e295.
- 31. Pearson MS, Bethony JM, Pickering DA, de Oliveira LM, Jariwala A, Santiago H, Miles AP, et al. An enzymatically inactivated hemoglobinase from Necator americanus induces neutralizing antibodies against multiple hookworm species and protects dogs against heterologous hookworm infection. Faseb J 2009;23:3007-3019.
- 32. Zhan B, Liu S, Perally S, Xue J, Fujiwara R, Brophy P, Xiao S, et al. Biochemical characterization and vaccine potential of a heme-binding glutathione transferase from the adult hookworm Ancylostoma caninum. Infect Immun 2005;73:6903-6911.
- 33. Zhan B, Perally S, Brophy PM, Xue J, Goud G, Liu S, Deumic V, et al. Molecular Cloning, Biochemical Characterization and Partial Protective Immunity of the Heme-binding Glutathione S-Transferases from the Human Hookworm Necator americanus. Infect Immun.
- 34. Asojo OA, Homma K, Sedlacek M, Ngamelue M, Goud GN, Zhan B, Deumic V, et al. X-ray structures of Na-GST-1 and Na-GST-2 two glutathione S-transferase from the human hookworm Necator americanus. BMC Struct Biol 2007;7:42.

- 35. van Rossum AJ, Jefferies JR, Rijsewijk FA, LaCourse EJ, Teesdale-Spittle P, Barrett J, Tait A, et al. Binding of hematin by a new class of glutathione transferase from the blood-feeding parasitic nematode Haemonchus contortus. Infect Immun 2004;72:2780-2790.
- 36. Schuller DJ, Liu Q, Kriksunov IA, Campbell AM, Barrett J, Brophy PM, Hao Q. Crystal structure of a new class of glutathione transferase from the model human hookworm nematode Heligmosomoides polygyrus. Proteins 2005;61:1024-1031.
- 37. Zhan B, Perally S, Brophy PM, Xue J, Goud G, Liu S, Deumic V, et al. Molecular cloning, biochemical characterization, and partial protective immunity of the heme-binding glutathione S-transferases from the human hookworm Necator americanus. Infect Immun 2010;78:1552-1563.
- 38. Xiao S, Zhan B, Xue J, Goud GN, Loukas A, Liu Y, Williamson A, et al. The evaluation of recombinant hookworm antigens as vaccines in hamsters (Mesocricetus auratus) challenged with human hookworm, Necator americanus. Exp Parasitol 2008;118:32-40.
- 39. Cody CL, Baraff LJ, Cherry JD, Marcy SM, Manclark CR. Nature and rates of adverse reactions associated with DTP and DT immunizations in infants and children. Pediatrics 1981;68:650-660.
- 40. Merck and Co. I. Recombivax HB® Product Insert. Whitehouse Station, NJ: Merck & Co., Inc., 2003.
- 41. Ribi E, Cantrell JL, Takayama K, Qureshi N, Peterson J, Ribi HO. Lipid A and immunotherapy. Rev Infect Dis 1984;6:567-572.
- 42. Ogutu BR, Apollo OJ, McKinney D, Okoth W, Siangla J, Dubovsky F, Tucker K, et al. Blood stage malaria vaccine eliciting high antigen-specific antibody concentrations confers no protection to young children in Western Kenya. PLoS One 2009;4:e4708.
- 43. Thera MA, Doumbo OK, Coulibaly D, Laurens MB, Kone AK, Guindo AB, Traore K, et al. Safety and immunogenicity of an AMA1 malaria vaccine in Malian children: results of a phase 1 randomized controlled trial. PLoS One 2010;5:e9041.
- 44. Sacarlal J, Aide P, Aponte JJ, Renom M, Leach A, Mandomando I, Lievens M, et al. Long-term safety and efficacy of the RTS,S/AS02A malaria vaccine in Mozambican children. J Infect Dis 2009;200:329-336.
- 45. Velez ID, Gilchrist K, Martinez S, Ramirez-Pineda JR, Ashman JA, Alves FP, Coler RN, et al. Safety and immunogenicity of a defined vaccine for the prevention of cutaneous leishmaniasis. Vaccine 2009;28:329-337.
- 46. Vandepapeliere P, Horsmans Y, Moris P, Van Mechelen M, Janssens M, Koutsoukos M, Van Belle P, et al. Vaccine adjuvant systems containing monophosphoryl lipid A and QS21 induce strong and persistent humoral and T cell responses against hepatitis B surface antigen in healthy adult volunteers. Vaccine 2008;26:1375-1386.
- 47. Paavonen J, Naud P, Salmeron J, Wheeler CM, Chow SN, Apter D, Kitchener H, et al. Efficacy of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine against cervical infection and precancer caused by oncogenic HPV types (PATRICIA): final analysis of a double-blind, randomised study in young women. Lancet 2009;374:301-314.
- 48. Konno R, Dobbelaere KO, Godeaux OO, Tamura S, Yoshikawa H. Immunogenicity, reactogenicity, and safety of human papillomavirus 16/18 AS04-adjuvanted vaccine in Japanese women: interim analysis of a phase II, double-blind, randomized controlled trial at month 7. Int J Gynecol Cancer 2009;19:905-911.
- 49. Behzad H, Huckriede AL, Haynes L, Gentleman B, Coyle K, Wilschut JC, Kollmann TR, et al. GLA-SE, a synthetic toll-like receptor 4 agonist, enhances T-cell responses to influenza vaccine in older adults. J Infect Dis 2012;205:466-473.
- 50. Hotez PJ, Bethony JM, Diemert DJ, Pearson M, Loukas A. Developing vaccines to combat hookworm infection and intestinal schistosomiasis. Nat Rev Microbiol 2010;8:814-826.

51. Treanor JJ, Essink B, Hull S, Reed S, Izikson R, Patriarca P, Goldenthal KL, et al. Evaluation of safety and immunogenicity of recombinant influenza hemagglutinin (H5/Indonesia/05/2005) formulated with and without a stable oil-in-water emulsion containing glucopyranosyl-lipid A (SE+GLA) adjuvant. Vaccine 2013;31:5760-5765.

# **SUPPLEMENTS/APPENDICES**

## **APPENDIX A: SCHEDULE OF EVENTS**

| Procedures | Blood<br>Volu<br>me | | | | | | | | | | | Study | / Day | 'S | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Pre<br>1 | 0 | 1 | 3<br>± 1 | 7<br>±1 | 14<br>±2 | 28<br>±4 | 56<br>±7 | 57 | 59<br>±1 | 63<br>±1 | 70<br>±2 | 84<br>±4 | 112<br>±14 | 113 | 115<br>±1 | 119<br>±1 | 126<br>±2 | 140<br>±4 | | | 380<br>±21 |
| Obtain Informed Consent | | Χ | | | | | | | | | | | | | | | | | | | | | |
| Complete History/Physical | | Х | | | | | | | | | | | | | | | | | | | | | |
| Interim Clinical Evaluation | | | Χ | Χ | Х | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Х | Χ | Χ | Х | Х | Х |
| AE/SAE/AESI Asessment | | | Χ | Χ | Х | Х | Х | Х | Х | Х | Χ | Х | Χ | Х | Х | Χ | Х | Х | Х | Χ | Х | Х | Х |
| Urine Dipstick | | Х | | | | | | | | | | | | | | | | | | | | | |
| Urine Pregnancy Test<br>(Females) | | Х | Х | | | | | | Х | | | | | | Х | | | | | | | | |
| HCV | | Х | | | | | | | | | | | | | | | | | | | | | |
| HBsAg | 10 mL | Х | | | | | | | | | | | | | | | | | | | | | |
| HIV | | Х | | | | | | | | | | | | | | | | | | | | | |
| Glucose (Random) | | Х | | | | | | | | | | | | | | | | | | | | | |
| ALT | 5 mL | Х | Х | | | | Х | | Х | | | | Χ | | Х | | | | Х | | | | |
| Creatinine | | Х | Χ | | | | Х | | Χ | | | | Х | | Χ | | | | Х | | | | |
| CBC <sup>2</sup> | 2 mL | Χ | Χ | | | | Χ | | Χ | | | | Χ | | Χ | | | | Χ | | | | |
| Serum and Plasma<br>Antibody Assays | 10 mL | Х | Х | | | х | Х | Х | Х | | | Х | Х | Х | X | | | Х | Х | Х | Х | Х | Х |
| Cellular Assays | 30 mL | | Χ | | | Χ | Χ | Х | Χ | | | Х | Х | Χ | Χ | | | Χ | Χ | Х | Χ | Χ | Х |
| Daily Blood<br>Volume (mL) | | 27 | 47 | | | 30 | 47 | 40 | 47 | | | 30 | 47 | 40 | 47 | | | 30 | 47 | 40 | 40 | 40 | 40 |
| Total Blood<br>Volume (mL) | | 27 | 74 | | | 114 | 161 | 201 | 248 | | | 288 | 335 | 375 | 422 | | | 462 | 509 | 549 | 589 | 629 | 669 |
| Stool Examination | | Х | | | | | | | | | | | | | | | | | | Х | | | Х |
| VACCINATIONS | | | 1 | | | | | | 2 | | | | | | 3 | | | | | | | | |

<sup>&</sup>lt;sup>1</sup>Completed within 90 days of first vaccination <sup>2</sup>CBC safety parameters include WBC, absolute neutrophil count, hemoglobin, and platelet count